CLINICAL TRIAL: NCT01721837
Title: Use of Pradaxa® (Dabigatran Etexilate) for Stroke Prevention in Patients With Nonvalvular Atrial Fibrillation and Mild to Moderate Renal Impairment
Brief Title: Dabigatran Etexilate for Stroke Prevention in Patients With Atrial Fibrillation and Mild to Moderate Renal Impairment
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1160.170
Record Dates: First submitted 2012-11-02; First posted 2012-11-06 (Estimated); Results first posted 2014-07-31 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-06

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Atrial fibrillation and mild to moderate renal impairment

SUMMARY:
Non-interventional, observational study of physicians' use of Dabigatran etexilate for stroke prevention in patients with atrial fibrillation and mild to moderate renal impairment

ELIGIBILITY:
Inclusion criteria:

* patients with atrial fibrillation foreseen for Pradaxa anticoagulation according to physician's decision for stroke prevention
* patients with mild or moderate renal impairment
* age >= 18 years at enrollment

Exclusion criteria:

- severe renal impairment (Creatinine Clearance < 30 ml/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients
Sampling Method: Non-Probability Sample
Enrollment: 4340 (Actual)
Dates: Start 2012-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1616):
- Germany (1616):
  - Boehringer Ingelheim Investigational Site 626, Aachen
  - Boehringer Ingelheim Investigational Site 627, Aachen
  - Boehringer Ingelheim Investigational Site 642, Aachen
  - Boehringer Ingelheim Investigational Site 643, Aachen
  - Boehringer Ingelheim Investigational Site 156, Aalen
  - Boehringer Ingelheim Investigational Site 159, Aalen
  - Boehringer Ingelheim Investigational Site 472, Aarbergen
  - Boehringer Ingelheim Investigational Site 830, Ahaus
  - Boehringer Ingelheim Investigational Site 834, Ahaus
  - Boehringer Ingelheim Investigational Site 853, Ahaus
  - Boehringer Ingelheim Investigational Site 858, Ahaus
  - Boehringer Ingelheim Investigational Site 842, Ahaus-Alstaette
  - Boehringer Ingelheim Investigational Site 1154, Ahrensburg
  - Boehringer Ingelheim Investigational Site 169, Aichtal
  - Boehringer Ingelheim Investigational Site 178, Aichtal
  - Boehringer Ingelheim Investigational Site 900, Albersloh
  - Boehringer Ingelheim Investigational Site 76, Albstadt
  - Boehringer Ingelheim Investigational Site 80, Albstadt
  - Boehringer Ingelheim Investigational Site 98, Albstadt
  - Boehringer Ingelheim Investigational Site 95, Albstadt-Ebingen
  - Boehringer Ingelheim Investigational Site 954, Alfeld
  - Boehringer Ingelheim Investigational Site 668, Alfter
  - Boehringer Ingelheim Investigational Site 211, Allersberg
  - Boehringer Ingelheim Investigational Site 473, Alpenrod
  - Boehringer Ingelheim Investigational Site 1246, Altenburg
  - Boehringer Ingelheim Investigational Site 1247, Altenburg
  - Boehringer Ingelheim Investigational Site 1268, Altenburg
  - Boehringer Ingelheim Investigational Site 1127, Altenholz
  - Boehringer Ingelheim Investigational Site 1161, Altenholz
  - Boehringer Ingelheim Investigational Site 543, Altenstadt
  - Boehringer Ingelheim Investigational Site 146, Altlußheim
  - Boehringer Ingelheim Investigational Site 225, Alzenau in Unterfranken
  - Boehringer Ingelheim Investigational Site 226, Alzenau in Unterfranken
  - Boehringer Ingelheim Investigational Site 228, Alzenau in Unterfranken
  - Boehringer Ingelheim Investigational Site 347, Amberg
  - Boehringer Ingelheim Investigational Site 350, Amberg
  - Boehringer Ingelheim Investigational Site 362, Amberg
  - Boehringer Ingelheim Investigational Site 1366, Anderbeck
  - Boehringer Ingelheim Investigational Site 1225, Apolda
  - Boehringer Ingelheim Investigational Site 1233, Apolda
  - Boehringer Ingelheim Investigational Site 1217, Arenshausen
  - Boehringer Ingelheim Investigational Site 818, Arnsberg
  - Boehringer Ingelheim Investigational Site 1222, Arnstadt
  - Boehringer Ingelheim Investigational Site 1224, Arnstadt
  - Boehringer Ingelheim Investigational Site 789, Attendorn
  - Boehringer Ingelheim Investigational Site 295, Attenkirchen
  - Boehringer Ingelheim Investigational Site 13, Au am Rhein
  - Boehringer Ingelheim Investigational Site 1262, Aue
  - Boehringer Ingelheim Investigational Site 302, Augsburg
  - Boehringer Ingelheim Investigational Site 303, Augsburg
  - Boehringer Ingelheim Investigational Site 306, Augsburg
  - Boehringer Ingelheim Investigational Site 315, Augsburg
  - Boehringer Ingelheim Investigational Site 326, Augsburg
  - Boehringer Ingelheim Investigational Site 327, Augsburg
  - Boehringer Ingelheim Investigational Site 276, Babensham
  - Boehringer Ingelheim Investigational Site 1074, Bad Bederkesa
  - Boehringer Ingelheim Investigational Site 1030, Bad Bentheim
  - Boehringer Ingelheim Investigational Site 478, Bad Breisig
  - Boehringer Ingelheim Investigational Site 1190, Bad Doberan
  - Boehringer Ingelheim Investigational Site 803, Bad Driburg
  - Boehringer Ingelheim Investigational Site 1267, Bad Elster
  - Boehringer Ingelheim Investigational Site 442, Bad Ems
  - Boehringer Ingelheim Investigational Site 443, Bad Ems
  - Boehringer Ingelheim Investigational Site 457, Bad Ems
  - Boehringer Ingelheim Investigational Site 137, Bad Friedrichshall
  - Boehringer Ingelheim Investigational Site 530, Bad Homburg v.d.H.
  - Boehringer Ingelheim Investigational Site 531, Bad Homburg v.d.H.
  - Boehringer Ingelheim Investigational Site 533, Bad Homburg v.d.H.
  - Boehringer Ingelheim Investigational Site 1250, Bad Klosterlausnitz
  - Boehringer Ingelheim Investigational Site 446, Bad Kreuznach
  - Boehringer Ingelheim Investigational Site 4, Bad Krozingen
  - Boehringer Ingelheim Investigational Site 1204, Bad Langensalza
  - Boehringer Ingelheim Investigational Site 932, Bad Lauterberg im Harz
  - Boehringer Ingelheim Investigational Site 934, Bad Lauterberg im Harz
  - Boehringer Ingelheim Investigational Site 937, Bad Lauterberg im Harz
  - Boehringer Ingelheim Investigational Site 680, Bad Münstereifel
  - Boehringer Ingelheim Investigational Site 453, Bad Nauheim
  - Boehringer Ingelheim Investigational Site 454, Bad Nauheim
  - Boehringer Ingelheim Investigational Site 528, Bad Nauheim
  - Boehringer Ingelheim Investigational Site 529, Bad Nauheim
  - Boehringer Ingelheim Investigational Site 1564, Bad Nenndorf
  - Boehringer Ingelheim Investigational Site 989, Bad Nenndorf
  - Boehringer Ingelheim Investigational Site 448, Bad Neuenahr
  - Boehringer Ingelheim Investigational Site 224, Bad Neustadt an der Saale
  - Boehringer Ingelheim Investigational Site 986, Bad Pyrmont
  - Boehringer Ingelheim Investigational Site 252, Bad Reichenhall
  - Boehringer Ingelheim Investigational Site 253, Bad Reichenhall
  - Boehringer Ingelheim Investigational Site 935, Bad Sachsa
  - Boehringer Ingelheim Investigational Site 936, Bad Sachsa
  - Boehringer Ingelheim Investigational Site 874, Bad Salzuflen
  - Boehringer Ingelheim Investigational Site 890, Bad Salzuflen
  - Boehringer Ingelheim Investigational Site 1207, Bad Salzungen
  - Boehringer Ingelheim Investigational Site 1219, Bad Salzungen
  - Boehringer Ingelheim Investigational Site 20, Bad Säckingen
  - Boehringer Ingelheim Investigational Site 87, Bad Schussenried
  - Boehringer Ingelheim Investigational Site 88, Bad Schussenried
  - Boehringer Ingelheim Investigational Site 1103, Bad Schwartau
  - Boehringer Ingelheim Investigational Site 1123, Bad Schwartau
  - Boehringer Ingelheim Investigational Site 532, Bad Soden am Taunus
  - Boehringer Ingelheim Investigational Site 1229, Bad Sulza
  - Boehringer Ingelheim Investigational Site 1582, Bad Tennstedt
  - Boehringer Ingelheim Investigational Site 1583, Bad Tennstedt
  - Boehringer Ingelheim Investigational Site 102, Bad Überkingen
  - Boehringer Ingelheim Investigational Site 78, Bad Waldsee
  - Boehringer Ingelheim Investigational Site 259, Bad Wiesee
  - Boehringer Ingelheim Investigational Site 235, Bad Wiessee
  - Boehringer Ingelheim Investigational Site 42, Bad Wildbad
  - Boehringer Ingelheim Investigational Site 68, Bad Wildbad
  - Boehringer Ingelheim Investigational Site 1375, Badel
  - Boehringer Ingelheim Investigational Site 3, Baden-Baden
  - Boehringer Ingelheim Investigational Site 961, Badenhausen
  - Boehringer Ingelheim Investigational Site 83, Baindt
  - Boehringer Ingelheim Investigational Site 84, Baindt
  - Boehringer Ingelheim Investigational Site 1488, Bamberg
  - Boehringer Ingelheim Investigational Site 1494, Bamberg
  - Boehringer Ingelheim Investigational Site 1592, Bamberg
  - Boehringer Ingelheim Investigational Site 1232, Barchfeld
  - Boehringer Ingelheim Investigational Site 1153, Bargteheide
  - Boehringer Ingelheim Investigational Site 1026, Barssel/Harkebruegge
  - Boehringer Ingelheim Investigational Site 1514, Barssel/Harkebruegge
  - Boehringer Ingelheim Investigational Site 1434, Baruth
  - Boehringer Ingelheim Investigational Site 1587, Bassum
  - Boehringer Ingelheim Investigational Site 971, Bassum
  - Boehringer Ingelheim Investigational Site 445, Baumholder
  - Boehringer Ingelheim Investigational Site 450, Baumholder
  - Boehringer Ingelheim Investigational Site 570, Baunatal
  - Boehringer Ingelheim Investigational Site 1437, Bautzen
  - Boehringer Ingelheim Investigational Site 1597, Bayreuth
  - Boehringer Ingelheim Investigational Site 378, Bayreuth
  - Boehringer Ingelheim Investigational Site 415, Bechhofen
  - Boehringer Ingelheim Investigational Site 883, Beckum
  - Boehringer Ingelheim Investigational Site 884, Beckum
  - Boehringer Ingelheim Investigational Site 1460, Beilrode
  - Boehringer Ingelheim Investigational Site 219, Bellngries
  - Boehringer Ingelheim Investigational Site 466, Bendorf
  - Boehringer Ingelheim Investigational Site 489, Bensheim
  - Boehringer Ingelheim Investigational Site 517, Bensheim
  - Boehringer Ingelheim Investigational Site 908, Berg. Gladbach
  - Boehringer Ingelheim Investigational Site 1195, Bergen
  - Boehringer Ingelheim Investigational Site 814, Bergkamen-Ruenthe
  - Boehringer Ingelheim Investigational Site 1143, Berlin
  - Boehringer Ingelheim Investigational Site 1270, Berlin
  - Boehringer Ingelheim Investigational Site 1271, Berlin
  - Boehringer Ingelheim Investigational Site 1277, Berlin
  - Boehringer Ingelheim Investigational Site 1278, Berlin
  - Boehringer Ingelheim Investigational Site 1279, Berlin
  - Boehringer Ingelheim Investigational Site 1280, Berlin
  - Boehringer Ingelheim Investigational Site 1281, Berlin
  - Boehringer Ingelheim Investigational Site 1282, Berlin
  - Boehringer Ingelheim Investigational Site 1285, Berlin
  - Boehringer Ingelheim Investigational Site 1304, Berlin
  - Boehringer Ingelheim Investigational Site 1305, Berlin
  - Boehringer Ingelheim Investigational Site 1306, Berlin
  - Boehringer Ingelheim Investigational Site 1307, Berlin
  - Boehringer Ingelheim Investigational Site 1309, Berlin
  - Boehringer Ingelheim Investigational Site 1310, Berlin
  - Boehringer Ingelheim Investigational Site 1311, Berlin
  - Boehringer Ingelheim Investigational Site 1312, Berlin
  - Boehringer Ingelheim Investigational Site 1315, Berlin
  - Boehringer Ingelheim Investigational Site 1316, Berlin
  - Boehringer Ingelheim Investigational Site 1318, Berlin
  - Boehringer Ingelheim Investigational Site 1319, Berlin
  - Boehringer Ingelheim Investigational Site 1320, Berlin
  - Boehringer Ingelheim Investigational Site 1321, Berlin
  - Boehringer Ingelheim Investigational Site 1322, Berlin
  - Boehringer Ingelheim Investigational Site 1323, Berlin
  - Boehringer Ingelheim Investigational Site 1325, Berlin
  - Boehringer Ingelheim Investigational Site 1326, Berlin
  - Boehringer Ingelheim Investigational Site 1328, Berlin
  - Boehringer Ingelheim Investigational Site 1329, Berlin
  - Boehringer Ingelheim Investigational Site 1330, Berlin
  - Boehringer Ingelheim Investigational Site 1331, Berlin
  - Boehringer Ingelheim Investigational Site 1336, Berlin
  - Boehringer Ingelheim Investigational Site 1338, Berlin
  - Boehringer Ingelheim Investigational Site 1377, Berlin
  - Boehringer Ingelheim Investigational Site 1382, Berlin
  - Boehringer Ingelheim Investigational Site 1384, Berlin
  - Boehringer Ingelheim Investigational Site 1385, Berlin
  - Boehringer Ingelheim Investigational Site 1386, Berlin
  - Boehringer Ingelheim Investigational Site 1387, Berlin
  - Boehringer Ingelheim Investigational Site 1388, Berlin
  - Boehringer Ingelheim Investigational Site 1389, Berlin
  - Boehringer Ingelheim Investigational Site 1390, Berlin
  - Boehringer Ingelheim Investigational Site 1406, Berlin
  - Boehringer Ingelheim Investigational Site 1407, Berlin
  - Boehringer Ingelheim Investigational Site 1408, Berlin
  - Boehringer Ingelheim Investigational Site 1540, Berlin
  - Boehringer Ingelheim Investigational Site 1541, Berlin
  - Boehringer Ingelheim Investigational Site 1542, Berlin
  - Boehringer Ingelheim Investigational Site 1543, Berlin
  - Boehringer Ingelheim Investigational Site 1544, Berlin
  - Boehringer Ingelheim Investigational Site 1545, Berlin
  - Boehringer Ingelheim Investigational Site 1546, Berlin
  - Boehringer Ingelheim Investigational Site 1547, Berlin
  - Boehringer Ingelheim Investigational Site 1549, Berlin
  - Boehringer Ingelheim Investigational Site 393, Berlin
  - Boehringer Ingelheim Investigational Site 1308, Bernau
  - Boehringer Ingelheim Investigational Site 1550, Bernau
  - Boehringer Ingelheim Investigational Site 1433, Bernsdorf
  - Boehringer Ingelheim Investigational Site 460, Beselich-Obertiefenbach
  - Boehringer Ingelheim Investigational Site 474, Beselich-Obertiefenbach
  - Boehringer Ingelheim Investigational Site 611, Bettingen
  - Boehringer Ingelheim Investigational Site 823, Beverungen
  - Boehringer Ingelheim Investigational Site 77, Biberach
  - Boehringer Ingelheim Investigational Site 512, Biblis
  - Boehringer Ingelheim Investigational Site 563, Biedenkopf
  - Boehringer Ingelheim Investigational Site 584, Biedenkopf
  - Boehringer Ingelheim Investigational Site 876, Bielefeld
  - Boehringer Ingelheim Investigational Site 901, Bielefeld
  - Boehringer Ingelheim Investigational Site 94, Bingen
  - Boehringer Ingelheim Investigational Site 1215, Bischofferode
  - Boehringer Ingelheim Investigational Site 504, Bischofsheim
  - Boehringer Ingelheim Investigational Site 1376, Bismark
  - Boehringer Ingelheim Investigational Site 1085, Bispingen
  - Boehringer Ingelheim Investigational Site 1370, Bitterfeld-Wolfen
  - Boehringer Ingelheim Investigational Site 1371, Bitterfeld-Wolfen
  - Boehringer Ingelheim Investigational Site 92, Blaubeuren Abbey
  - Boehringer Ingelheim Investigational Site 1580, Bleicherode
  - Boehringer Ingelheim Investigational Site 896, Blomberg
  - Boehringer Ingelheim Investigational Site 57, Blumberg
  - Boehringer Ingelheim Investigational Site 1420, Bobritzsch
  - Boehringer Ingelheim Investigational Site 769, Bochum
  - Boehringer Ingelheim Investigational Site 771, Bochum
  - Boehringer Ingelheim Investigational Site 773, Bochum
  - Boehringer Ingelheim Investigational Site 775, Bochum
  - Boehringer Ingelheim Investigational Site 777, Bochum
  - Boehringer Ingelheim Investigational Site 778, Bochum
  - Boehringer Ingelheim Investigational Site 779, Bochum
  - Boehringer Ingelheim Investigational Site 780, Bochum
  - Boehringer Ingelheim Investigational Site 339, Bodenkirchen
  - Boehringer Ingelheim Investigational Site 682, Bonn
  - Boehringer Ingelheim Investigational Site 41, Bonndorf
  - Boehringer Ingelheim Investigational Site 55, Bonndorf
  - Boehringer Ingelheim Investigational Site 1137, Boostedt
  - Boehringer Ingelheim Investigational Site 158, Bopfingen
  - Boehringer Ingelheim Investigational Site 1162, Bordesholm
  - Boehringer Ingelheim Investigational Site 899, Borgholzhausen
  - Boehringer Ingelheim Investigational Site 844, Borken
  - Boehringer Ingelheim Investigational Site 1476, Borna
  - Boehringer Ingelheim Investigational Site 838, Bottrop
  - Boehringer Ingelheim Investigational Site 852, Bottrop
  - Boehringer Ingelheim Investigational Site 962, Bovenden-Reyershausen
  - Boehringer Ingelheim Investigational Site 1572, Böblingen
  - Boehringer Ingelheim Investigational Site 48, Böblingen
  - Boehringer Ingelheim Investigational Site 51, Böblingen
  - Boehringer Ingelheim Investigational Site 1457, Böhlen
  - Boehringer Ingelheim Investigational Site 1010, Brake
  - Boehringer Ingelheim Investigational Site 1023, Brake
  - Boehringer Ingelheim Investigational Site 1038, Bramsche
  - Boehringer Ingelheim Investigational Site 1456, Braunsbedra
  - Boehringer Ingelheim Investigational Site 940, Braunschweig
  - Boehringer Ingelheim Investigational Site 941, Braunschweig
  - Boehringer Ingelheim Investigational Site 943, Braunschweig
  - Boehringer Ingelheim Investigational Site 949, Braunschweig
  - Boehringer Ingelheim Investigational Site 54, Bräunlingen
  - Boehringer Ingelheim Investigational Site 1496, Breitenguessbach
  - Boehringer Ingelheim Investigational Site 1053, Bremen
  - Boehringer Ingelheim Investigational Site 1061, Bremen
  - Boehringer Ingelheim Investigational Site 1062, Bremen
  - Boehringer Ingelheim Investigational Site 1063, Bremen
  - Boehringer Ingelheim Investigational Site 1064, Bremen
  - Boehringer Ingelheim Investigational Site 1065, Bremen
  - Boehringer Ingelheim Investigational Site 1066, Bremen
  - Boehringer Ingelheim Investigational Site 1067, Bremen
  - Boehringer Ingelheim Investigational Site 1068, Bremen
  - Boehringer Ingelheim Investigational Site 1069, Bremen
  - Boehringer Ingelheim Investigational Site 1045, Bremerhaven
  - Boehringer Ingelheim Investigational Site 1046, Bremerhaven
  - Boehringer Ingelheim Investigational Site 1048, Bremerhaven
  - Boehringer Ingelheim Investigational Site 1079, Bremerhaven
  - Boehringer Ingelheim Investigational Site 1050, Bremervörde
  - Boehringer Ingelheim Investigational Site 143, Bretten
  - Boehringer Ingelheim Investigational Site 1611, Bretten
  - Boehringer Ingelheim Investigational Site 806, Brilon
  - Boehringer Ingelheim Investigational Site 431, Bruchweiler-Baerenbach
  - Boehringer Ingelheim Investigational Site 363, Bruck
  - Boehringer Ingelheim Investigational Site 337, Buchbach
  - Boehringer Ingelheim Investigational Site 338, Buchbach
  - Boehringer Ingelheim Investigational Site 1051, Buchholz
  - Boehringer Ingelheim Investigational Site 1083, Buchholz
  - Boehringer Ingelheim Investigational Site 1335, Buckow
  - Boehringer Ingelheim Investigational Site 1294, Burg
  - Boehringer Ingelheim Investigational Site 980, Burgdorf, Hanover
  - Boehringer Ingelheim Investigational Site 985, Burgdorf, Hanover
  - Boehringer Ingelheim Investigational Site 1432, Burgneudorf
  - Boehringer Ingelheim Investigational Site 557, Butzbach
  - Boehringer Ingelheim Investigational Site 1145, Büchen
  - Boehringer Ingelheim Investigational Site 1146, Büchen
  - Boehringer Ingelheim Investigational Site 1500, Büchen
  - Boehringer Ingelheim Investigational Site 1519, Büchen
  - Boehringer Ingelheim Investigational Site 968, Bückeburg
  - Boehringer Ingelheim Investigational Site 878, Bünde
  - Boehringer Ingelheim Investigational Site 828, Büren
  - Boehringer Ingelheim Investigational Site 800, Castrop-Rauxel
  - Boehringer Ingelheim Investigational Site 810, Castrop-Rauxel
  - Boehringer Ingelheim Investigational Site 812, Castrop-Rauxel
  - Boehringer Ingelheim Investigational Site 824, Castrop-Rauxel
  - Boehringer Ingelheim Investigational Site 1239, Chemnitz
  - Boehringer Ingelheim Investigational Site 1240, Chemnitz
  - Boehringer Ingelheim Investigational Site 1241, Chemnitz
  - Boehringer Ingelheim Investigational Site 1242, Chemnitz
  - Boehringer Ingelheim Investigational Site 1253, Chemnitz
  - Boehringer Ingelheim Investigational Site 1256, Chemnitz
  - Boehringer Ingelheim Investigational Site 1257, Chemnitz
  - Boehringer Ingelheim Investigational Site 1258, Chemnitz
  - Boehringer Ingelheim Investigational Site 1259, Chemnitz
  - Boehringer Ingelheim Investigational Site 1260, Chemnitz
  - Boehringer Ingelheim Investigational Site 409, Coburg
  - Boehringer Ingelheim Investigational Site 477, Cochem
  - Boehringer Ingelheim Investigational Site 629, Cologne
  - Boehringer Ingelheim Investigational Site 630, Cologne
  - Boehringer Ingelheim Investigational Site 631, Cologne
  - Boehringer Ingelheim Investigational Site 633, Cologne
  - Boehringer Ingelheim Investigational Site 634, Cologne
  - Boehringer Ingelheim Investigational Site 635, Cologne
  - Boehringer Ingelheim Investigational Site 646, Cologne
  - Boehringer Ingelheim Investigational Site 647, Cologne
  - Boehringer Ingelheim Investigational Site 651, Cologne
  - Boehringer Ingelheim Investigational Site 655, Cologne
  - Boehringer Ingelheim Investigational Site 656, Cologne
  - Boehringer Ingelheim Investigational Site 660, Cologne
  - Boehringer Ingelheim Investigational Site 661, Cologne
  - Boehringer Ingelheim Investigational Site 662, Cologne
  - Boehringer Ingelheim Investigational Site 666, Cologne
  - Boehringer Ingelheim Investigational Site 670, Cologne
  - Boehringer Ingelheim Investigational Site 673, Cologne
  - Boehringer Ingelheim Investigational Site 674, Cologne
  - Boehringer Ingelheim Investigational Site 1354, Coswig
  - Boehringer Ingelheim Investigational Site 1292, Cottbus
  - Boehringer Ingelheim Investigational Site 1296, Crinitz
  - Boehringer Ingelheim Investigational Site 296, Dachau
  - Boehringer Ingelheim Investigational Site 300, Dachau
  - Boehringer Ingelheim Investigational Site 1192, Dargun
  - Boehringer Ingelheim Investigational Site 488, Darmstadt
  - Boehringer Ingelheim Investigational Site 490, Darmstadt
  - Boehringer Ingelheim Investigational Site 516, Darmstadt
  - Boehringer Ingelheim Investigational Site 593, Dautphetal
  - Boehringer Ingelheim Investigational Site 354, Deggendorf
  - Boehringer Ingelheim Investigational Site 1466, Delitzsch
  - Boehringer Ingelheim Investigational Site 1599, Delitzsch
  - Boehringer Ingelheim Investigational Site 1194, Demmin
  - Boehringer Ingelheim Investigational Site 1356, Dessau
  - Boehringer Ingelheim Investigational Site 893, Detmold
  - Boehringer Ingelheim Investigational Site 526, Dieburg
  - Boehringer Ingelheim Investigational Site 527, Dieburg
  - Boehringer Ingelheim Investigational Site 999, Diepenau
  - Boehringer Ingelheim Investigational Site 586, Dietzhoelztal
  - Boehringer Ingelheim Investigational Site 238, Dießen
  - Boehringer Ingelheim Investigational Site 599, Dillingen/Saar
  - Boehringer Ingelheim Investigational Site 198, Dinkelsbühl
  - Boehringer Ingelheim Investigational Site 213, Dinkelsbühl
  - Boehringer Ingelheim Investigational Site 223, Dinkelsbühl
  - Boehringer Ingelheim Investigational Site 1028, Dinklage
  - Boehringer Ingelheim Investigational Site 725, Dinslaken
  - Boehringer Ingelheim Investigational Site 760, Dinslaken-Averbruch
  - Boehringer Ingelheim Investigational Site 405, Doerfles-Esbach
  - Boehringer Ingelheim Investigational Site 21, Dogern
  - Boehringer Ingelheim Investigational Site 700, Dormagen
  - Boehringer Ingelheim Investigational Site 638, Dortmund
  - Boehringer Ingelheim Investigational Site 641, Dortmund
  - Boehringer Ingelheim Investigational Site 795, Dortmund
  - Boehringer Ingelheim Investigational Site 796, Dortmund
  - Boehringer Ingelheim Investigational Site 797, Dortmund
  - Boehringer Ingelheim Investigational Site 798, Dortmund
  - Boehringer Ingelheim Investigational Site 799, Dortmund
  - Boehringer Ingelheim Investigational Site 801, Dortmund
  - Boehringer Ingelheim Investigational Site 802, Dortmund
  - Boehringer Ingelheim Investigational Site 809, Dortmund
  - Boehringer Ingelheim Investigational Site 825, Dortmund
  - Boehringer Ingelheim Investigational Site 550, Dreieich
  - Boehringer Ingelheim Investigational Site 554, Dreieich
  - Boehringer Ingelheim Investigational Site 552, Dreieich-Dreieichenhain
  - Boehringer Ingelheim Investigational Site 1410, Dresden
  - Boehringer Ingelheim Investigational Site 1411, Dresden
  - Boehringer Ingelheim Investigational Site 1426, Dresden
  - Boehringer Ingelheim Investigational Site 1427, Dresden
  - Boehringer Ingelheim Investigational Site 1429, Dresden
  - Boehringer Ingelheim Investigational Site 1430, Dresden
  - Boehringer Ingelheim Investigational Site 1431, Dresden
  - Boehringer Ingelheim Investigational Site 1441, Dresden
  - Boehringer Ingelheim Investigational Site 1442, Dresden
  - Boehringer Ingelheim Investigational Site 1443, Dresden
  - Boehringer Ingelheim Investigational Site 588, Driedorf
  - Boehringer Ingelheim Investigational Site 1093, Drochtersen
  - Boehringer Ingelheim Investigational Site 1094, Drochtersen
  - Boehringer Ingelheim Investigational Site 427, Dudenhofen
  - Boehringer Ingelheim Investigational Site 729, Duisburg
  - Boehringer Ingelheim Investigational Site 730, Duisburg
  - Boehringer Ingelheim Investigational Site 731, Duisburg
  - Boehringer Ingelheim Investigational Site 736, Duisburg
  - Boehringer Ingelheim Investigational Site 738, Duisburg
  - Boehringer Ingelheim Investigational Site 739, Duisburg
  - Boehringer Ingelheim Investigational Site 740, Duisburg
  - Boehringer Ingelheim Investigational Site 741, Duisburg
  - Boehringer Ingelheim Investigational Site 233, Durach
  - Boehringer Ingelheim Investigational Site 34, Durmersheim
  - Boehringer Ingelheim Investigational Site 1596, Düsseldorf
  - Boehringer Ingelheim Investigational Site 689, Düsseldorf
  - Boehringer Ingelheim Investigational Site 692, Düsseldorf
  - Boehringer Ingelheim Investigational Site 693, Düsseldorf
  - Boehringer Ingelheim Investigational Site 694, Düsseldorf
  - Boehringer Ingelheim Investigational Site 695, Düsseldorf
  - Boehringer Ingelheim Investigational Site 697, Düsseldorf
  - Boehringer Ingelheim Investigational Site 698, Düsseldorf
  - Boehringer Ingelheim Investigational Site 715, Düsseldorf
  - Boehringer Ingelheim Investigational Site 716, Düsseldorf
  - Boehringer Ingelheim Investigational Site 717, Düsseldorf
  - Boehringer Ingelheim Investigational Site 906, Düsseldorf
  - Boehringer Ingelheim Investigational Site 917, Düsseldorf
  - Boehringer Ingelheim Investigational Site 919, Düsseldorf
  - Boehringer Ingelheim Investigational Site 918, Düsseldorf-Benrath
  - Boehringer Ingelheim Investigational Site 1213, Ebeleben
  - Boehringer Ingelheim Investigational Site 964, Ebergötzen
  - Boehringer Ingelheim Investigational Site 580, Ebersburg-Schmalnau
  - Boehringer Ingelheim Investigational Site 1106, Eckernförde
  - Boehringer Ingelheim Investigational Site 1116, Eckernförde
  - Boehringer Ingelheim Investigational Site 1014, Edewecht
  - Boehringer Ingelheim Investigational Site 275, Edling
  - Boehringer Ingelheim Investigational Site 19, Efringen-Kirchen
  - Boehringer Ingelheim Investigational Site 86, Ehingen
  - Boehringer Ingelheim Investigational Site 26, Ehrenkirchen
  - Boehringer Ingelheim Investigational Site 535, Ehringshausen
  - Boehringer Ingelheim Investigational Site 200, Eichstätt
  - Boehringer Ingelheim Investigational Site 1482, Eilenburg
  - Boehringer Ingelheim Investigational Site 963, Einbeck
  - Boehringer Ingelheim Investigational Site 1303, Eisenhüttenstadt
  - Boehringer Ingelheim Investigational Site 154, Ellwangen/Jagst
  - Boehringer Ingelheim Investigational Site 1272, Elsterwerda
  - Boehringer Ingelheim Investigational Site 1274, Elsterwerda
  - Boehringer Ingelheim Investigational Site 1301, Elsterwerda
  - Boehringer Ingelheim Investigational Site 471, Elz
  - Boehringer Ingelheim Investigational Site 675, Engelskirchen-Ruenderoth
  - Boehringer Ingelheim Investigational Site 881, Ennigerloh-Ostenfelde
  - Boehringer Ingelheim Investigational Site 615, Eppelborn
  - Boehringer Ingelheim Investigational Site 140, Eppingen
  - Boehringer Ingelheim Investigational Site 1612, Eppingen
  - Boehringer Ingelheim Investigational Site 1134, Erfde
  - Boehringer Ingelheim Investigational Site 684, Erftstadt
  - Boehringer Ingelheim Investigational Site 686, Erftstadt
  - Boehringer Ingelheim Investigational Site 1212, Erfurt
  - Boehringer Ingelheim Investigational Site 1614, Erkelenz
  - Boehringer Ingelheim Investigational Site 654, Erkelenz
  - Boehringer Ingelheim Investigational Site 189, Erlangen
  - Boehringer Ingelheim Investigational Site 190, Erlangen
  - Boehringer Ingelheim Investigational Site 192, Erlangen
  - Boehringer Ingelheim Investigational Site 193, Erlangen
  - Boehringer Ingelheim Investigational Site 194, Erlangen
  - Boehringer Ingelheim Investigational Site 212, Erlangen
  - Boehringer Ingelheim Investigational Site 220, Erlangen
  - Boehringer Ingelheim Investigational Site 221, Erlangen
  - Boehringer Ingelheim Investigational Site 132, Erligheim
  - Boehringer Ingelheim Investigational Site 534, Eschborn
  - Boehringer Ingelheim Investigational Site 567, Eschwege
  - Boehringer Ingelheim Investigational Site 625, Eschweiler
  - Boehringer Ingelheim Investigational Site 898, Espelkamp
  - Boehringer Ingelheim Investigational Site 726, Essen
  - Boehringer Ingelheim Investigational Site 727, Essen
  - Boehringer Ingelheim Investigational Site 737, Essen
  - Boehringer Ingelheim Investigational Site 743, Essen
  - Boehringer Ingelheim Investigational Site 744, Essen
  - Boehringer Ingelheim Investigational Site 745, Essen
  - Boehringer Ingelheim Investigational Site 746, Essen
  - Boehringer Ingelheim Investigational Site 747, Essen
  - Boehringer Ingelheim Investigational Site 748, Essen
  - Boehringer Ingelheim Investigational Site 749, Essen
  - Boehringer Ingelheim Investigational Site 750, Essen
  - Boehringer Ingelheim Investigational Site 751, Essen
  - Boehringer Ingelheim Investigational Site 752, Essen
  - Boehringer Ingelheim Investigational Site 148, Esslingen am Neckar
  - Boehringer Ingelheim Investigational Site 36, Ettlingen
  - Boehringer Ingelheim Investigational Site 683, Euskirchen
  - Boehringer Ingelheim Investigational Site 1121, Eutin
  - Boehringer Ingelheim Investigational Site 1615, Eutin
  - Boehringer Ingelheim Investigational Site 1396, Falkensee
  - Boehringer Ingelheim Investigational Site 979, Faßberg
  - Boehringer Ingelheim Investigational Site 573, Felsberg-Gensungen
  - Boehringer Ingelheim Investigational Site 1104, Flensburg
  - Boehringer Ingelheim Investigational Site 1105, Flensburg
  - Boehringer Ingelheim Investigational Site 1107, Flensburg
  - Boehringer Ingelheim Investigational Site 1130, Flensburg
  - Boehringer Ingelheim Investigational Site 1133, Flensburg
  - Boehringer Ingelheim Investigational Site 547, Florstadt / Staden
  - Boehringer Ingelheim Investigational Site 1415, Flöha
  - Boehringer Ingelheim Investigational Site 1489, Forchheim
  - Boehringer Ingelheim Investigational Site 1490, Forchheim
  - Boehringer Ingelheim Investigational Site 585, Frankenberg
  - Boehringer Ingelheim Investigational Site 518, Frankfurt
  - Boehringer Ingelheim Investigational Site 522, Frankfurt
  - Boehringer Ingelheim Investigational Site 524, Frankfurt
  - Boehringer Ingelheim Investigational Site 1275, Frankfurt (Oder)
  - Boehringer Ingelheim Investigational Site 1283, Frankfurt (Oder)
  - Boehringer Ingelheim Investigational Site 1284, Frankfurt (Oder)
  - Boehringer Ingelheim Investigational Site 548, Frankfurt am Main
  - Boehringer Ingelheim Investigational Site 521, Frankfurt/M.
  - Boehringer Ingelheim Investigational Site 549, Frankfurt/M.
  - Boehringer Ingelheim Investigational Site 637, Frechen
  - Boehringer Ingelheim Investigational Site 1414, Freiberg
  - Boehringer Ingelheim Investigational Site 1425, Freiberg
  - Boehringer Ingelheim Investigational Site 1510, Freiburg im Breisgau
  - Boehringer Ingelheim Investigational Site 1, Freiburg im Breisgau
  - Boehringer Ingelheim Investigational Site 24, Freiburg im Breisgau
  - Boehringer Ingelheim Investigational Site 25, Freiburg im Breisgau
  - Boehringer Ingelheim Investigational Site 6, Freiburg im Breisgau
  - Boehringer Ingelheim Investigational Site 7, Freiburg im Breisgau
  - Boehringer Ingelheim Investigational Site 434, Freinsheim
  - Boehringer Ingelheim Investigational Site 292, Freising
  - Boehringer Ingelheim Investigational Site 1422, Freital
  - Boehringer Ingelheim Investigational Site 201, Fremdingen
  - Boehringer Ingelheim Investigational Site 380, Frensdorf
  - Boehringer Ingelheim Investigational Site 104, Friedrichshafen
  - Boehringer Ingelheim Investigational Site 106, Friedrichshafen
  - Boehringer Ingelheim Investigational Site 1556, Fritzlar
  - Boehringer Ingelheim Investigational Site 559, Fritzlar
  - Boehringer Ingelheim Investigational Site 807, Fröndenberg
  - Boehringer Ingelheim Investigational Site 820, Fröndenberg
  - Boehringer Ingelheim Investigational Site 822, Fröndenberg
  - Boehringer Ingelheim Investigational Site 340, Fuerstenfeldbruck-Aich
  - Boehringer Ingelheim Investigational Site 569, Fulda
  - Boehringer Ingelheim Investigational Site 342, Fürstenfeldbruck
  - Boehringer Ingelheim Investigational Site 1288, Fürstenwalde
  - Boehringer Ingelheim Investigational Site 1289, Fürstenwalde
  - Boehringer Ingelheim Investigational Site 377, Fürth
  - Boehringer Ingelheim Investigational Site 371, Gangkofen
  - Boehringer Ingelheim Investigational Site 323, Garching
  - Boehringer Ingelheim Investigational Site 1374, Gardelegen
  - Boehringer Ingelheim Investigational Site 237, Garmisch-Partenkirchen
  - Boehringer Ingelheim Investigational Site 248, Garmisch-Patenkirchen
  - Boehringer Ingelheim Investigational Site 556, Gedern-Wenings
  - Boehringer Ingelheim Investigational Site 1025, Geeste
  - Boehringer Ingelheim Investigational Site 1155, Geesthacht
  - Boehringer Ingelheim Investigational Site 837, Geisenkirchen-Buer
  - Boehringer Ingelheim Investigational Site 81, Geislingen/Steige
  - Boehringer Ingelheim Investigational Site 93, Geislingen/Steige
  - Boehringer Ingelheim Investigational Site 836, Gelsenkirchen
  - Boehringer Ingelheim Investigational Site 840, Gelsenkirchen
  - Boehringer Ingelheim Investigational Site 843, Gelsenkirchen
  - Boehringer Ingelheim Investigational Site 859, Gelsenkirchen
  - Boehringer Ingelheim Investigational Site 862, Gelsenkirchen
  - Boehringer Ingelheim Investigational Site 863, Gelsenkirchen
  - Boehringer Ingelheim Investigational Site 864, Gelsenkirchen
  - Boehringer Ingelheim Investigational Site 865, Gelsenkirchen
  - Boehringer Ingelheim Investigational Site 499, Gensingen
  - Boehringer Ingelheim Investigational Site 1339, Genthin
  - Boehringer Ingelheim Investigational Site 1340, Genthin
  - Boehringer Ingelheim Investigational Site 1235, Gera
  - Boehringer Ingelheim Investigational Site 1236, Gera
  - Boehringer Ingelheim Investigational Site 1237, Gera
  - Boehringer Ingelheim Investigational Site 264, Geretsried
  - Boehringer Ingelheim Investigational Site 40, Gerlingen
  - Boehringer Ingelheim Investigational Site 420, Germersheim
  - Boehringer Ingelheim Investigational Site 592, Gersfeld
  - Boehringer Ingelheim Investigational Site 91, Gerstetten
  - Boehringer Ingelheim Investigational Site 79, Giengen an der Brenz
  - Boehringer Ingelheim Investigational Site 1589, Giessen
  - Boehringer Ingelheim Investigational Site 1590, Giessen
  - Boehringer Ingelheim Investigational Site 560, Giessen
  - Boehringer Ingelheim Investigational Site 561, Giessen
  - Boehringer Ingelheim Investigational Site 942, Gifhorn
  - Boehringer Ingelheim Investigational Site 246, Gilching
  - Boehringer Ingelheim Investigational Site 1538, Glienicke/Glienicker Spitze
  - Boehringer Ingelheim Investigational Site 1539, Glienicke/Glienicker Spitze
  - Boehringer Ingelheim Investigational Site 1392, Glindow
  - Boehringer Ingelheim Investigational Site 1136, Glücksburg
  - Boehringer Ingelheim Investigational Site 966, Goettingen-Weende
  - Boehringer Ingelheim Investigational Site 1186, Goldberg
  - Boehringer Ingelheim Investigational Site 142, Gondelsheim
  - Boehringer Ingelheim Investigational Site 1417, Görlitz
  - Boehringer Ingelheim Investigational Site 1418, Görlitz
  - Boehringer Ingelheim Investigational Site 1439, Görlitz
  - Boehringer Ingelheim Investigational Site 205, Grafenrheinfeld
  - Boehringer Ingelheim Investigational Site 269, Gräfelfing
  - Boehringer Ingelheim Investigational Site 1461, Gräfenhainichen
  - Boehringer Ingelheim Investigational Site 1511, Grenzach-Wyhlen
  - Boehringer Ingelheim Investigational Site 511, Griesheim
  - Boehringer Ingelheim Investigational Site 1196, Grimmen
  - Boehringer Ingelheim Investigational Site 1125, Groß Grönau
  - Boehringer Ingelheim Investigational Site 551, Groß-Zimmern
  - Boehringer Ingelheim Investigational Site 456, Großmaischeid
  - Boehringer Ingelheim Investigational Site 603, Großrosseln
  - Boehringer Ingelheim Investigational Site 1502, Gröden
  - Boehringer Ingelheim Investigational Site 1526, Gröden
  - Boehringer Ingelheim Investigational Site 418, Grünstadt
  - Boehringer Ingelheim Investigational Site 185, Gschwend
  - Boehringer Ingelheim Investigational Site 659, Gummersbach
  - Boehringer Ingelheim Investigational Site 18, Gundelfingen
  - Boehringer Ingelheim Investigational Site 304, Günzburg
  - Boehringer Ingelheim Investigational Site 886, Gütersloh
  - Boehringer Ingelheim Investigational Site 887, Gütersloh
  - Boehringer Ingelheim Investigational Site 891, Gütersloh
  - Boehringer Ingelheim Investigational Site 903, Haan
  - Boehringer Ingelheim Investigational Site 914, Haan
  - Boehringer Ingelheim Investigational Site 273, Haar
  - Boehringer Ingelheim Investigational Site 444, Hachenburg
  - Boehringer Ingelheim Investigational Site 476, Hadamar
  - Boehringer Ingelheim Investigational Site 761, Hagen
  - Boehringer Ingelheim Investigational Site 762, Hagen
  - Boehringer Ingelheim Investigational Site 768, Hagen
  - Boehringer Ingelheim Investigational Site 781, Hagen
  - Boehringer Ingelheim Investigational Site 782, Hagen
  - Boehringer Ingelheim Investigational Site 783, Hagen
  - Boehringer Ingelheim Investigational Site 785, Hagen
  - Boehringer Ingelheim Investigational Site 786, Hagen
  - Boehringer Ingelheim Investigational Site 1522, Haibach
  - Boehringer Ingelheim Investigational Site 209, Haibach
  - Boehringer Ingelheim Investigational Site 1346, Halberstadt
  - Boehringer Ingelheim Investigational Site 1368, Halberstadt
  - Boehringer Ingelheim Investigational Site 1349, Haldensleben I
  - Boehringer Ingelheim Investigational Site 293, Hallbergmoos
  - Boehringer Ingelheim Investigational Site 1350, Halle
  - Boehringer Ingelheim Investigational Site 1351, Halle
  - Boehringer Ingelheim Investigational Site 1352, Halle
  - Boehringer Ingelheim Investigational Site 1355, Halle
  - Boehringer Ingelheim Investigational Site 1357, Halle
  - Boehringer Ingelheim Investigational Site 1358, Halle
  - Boehringer Ingelheim Investigational Site 1373, Halle
  - Boehringer Ingelheim Investigational Site 866, Halle
  - Boehringer Ingelheim Investigational Site 867, Halle
  - Boehringer Ingelheim Investigational Site 868, Halle
  - Boehringer Ingelheim Investigational Site 882, Halle
  - Boehringer Ingelheim Investigational Site 1495, Hallstadt
  - Boehringer Ingelheim Investigational Site 1054, Hamburg
  - Boehringer Ingelheim Investigational Site 1055, Hamburg
  - Boehringer Ingelheim Investigational Site 1056, Hamburg
  - Boehringer Ingelheim Investigational Site 1057, Hamburg
  - Boehringer Ingelheim Investigational Site 1058, Hamburg
  - Boehringer Ingelheim Investigational Site 1059, Hamburg
  - Boehringer Ingelheim Investigational Site 1090, Hamburg
  - Boehringer Ingelheim Investigational Site 1091, Hamburg
  - Boehringer Ingelheim Investigational Site 1092, Hamburg
  - Boehringer Ingelheim Investigational Site 1095, Hamburg
  - Boehringer Ingelheim Investigational Site 1096, Hamburg
  - Boehringer Ingelheim Investigational Site 1097, Hamburg
  - Boehringer Ingelheim Investigational Site 1098, Hamburg
  - Boehringer Ingelheim Investigational Site 1099, Hamburg
  - Boehringer Ingelheim Investigational Site 1108, Hamburg
  - Boehringer Ingelheim Investigational Site 1109, Hamburg
  - Boehringer Ingelheim Investigational Site 1110, Hamburg
  - Boehringer Ingelheim Investigational Site 1111, Hamburg
  - Boehringer Ingelheim Investigational Site 1118, Hamburg
  - Boehringer Ingelheim Investigational Site 1119, Hamburg
  - Boehringer Ingelheim Investigational Site 1147, Hamburg
  - Boehringer Ingelheim Investigational Site 1148, Hamburg
  - Boehringer Ingelheim Investigational Site 1149, Hamburg
  - Boehringer Ingelheim Investigational Site 1150, Hamburg
  - Boehringer Ingelheim Investigational Site 1156, Hamburg
  - Boehringer Ingelheim Investigational Site 1157, Hamburg
  - Boehringer Ingelheim Investigational Site 1163, Hamburg
  - Boehringer Ingelheim Investigational Site 1164, Hamburg
  - Boehringer Ingelheim Investigational Site 1168, Hamburg
  - Boehringer Ingelheim Investigational Site 1170, Hamburg
  - Boehringer Ingelheim Investigational Site 1506, Hamburg
  - Boehringer Ingelheim Investigational Site 1507, Hamburg
  - Boehringer Ingelheim Investigational Site 1523, Hamburg
  - Boehringer Ingelheim Investigational Site 1598, Hamburg
  - Boehringer Ingelheim Investigational Site 1152, Hamburg-Bergstedt
  - Boehringer Ingelheim Investigational Site 1501, Hamburg-Bergstedt
  - Boehringer Ingelheim Investigational Site 987, Hamelin
  - Boehringer Ingelheim Investigational Site 794, Hamm
  - Boehringer Ingelheim Investigational Site 816, Hamm
  - Boehringer Ingelheim Investigational Site 821, Hamm
  - Boehringer Ingelheim Investigational Site 227, Hammelburg
  - Boehringer Ingelheim Investigational Site 542, Hanau
  - Boehringer Ingelheim Investigational Site 546, Hanau
  - Boehringer Ingelheim Investigational Site 544, Hanau/M.
  - Boehringer Ingelheim Investigational Site 1002, Hanover
  - Boehringer Ingelheim Investigational Site 977, Hanover
  - Boehringer Ingelheim Investigational Site 981, Hanover
  - Boehringer Ingelheim Investigational Site 1052, Hanstedt
  - Boehringer Ingelheim Investigational Site 1089, Hanstedt
  - Boehringer Ingelheim Investigational Site 871, Harsewinkel
  - Boehringer Ingelheim Investigational Site 1024, Haselünne
  - Boehringer Ingelheim Investigational Site 241, Hausham
  - Boehringer Ingelheim Investigational Site 847, Havixbeck
  - Boehringer Ingelheim Investigational Site 413, Haßloch
  - Boehringer Ingelheim Investigational Site 436, Haßloch
  - Boehringer Ingelheim Investigational Site 129, Heddesheim
  - Boehringer Ingelheim Investigational Site 108, Heidelberg
  - Boehringer Ingelheim Investigational Site 113, Heidelberg
  - Boehringer Ingelheim Investigational Site 117, Heidelberg
  - Boehringer Ingelheim Investigational Site 118, Heidelberg
  - Boehringer Ingelheim Investigational Site 122, Heidelberg
  - Boehringer Ingelheim Investigational Site 127, Heidelberg
  - Boehringer Ingelheim Investigational Site 128, Heidelberg (Handschuhsheim)
  - Boehringer Ingelheim Investigational Site 72, Heidenheim
  - Boehringer Ingelheim Investigational Site 1581, Heilbad Heiligenstadt
  - Boehringer Ingelheim Investigational Site 120, Heilbronn
  - Boehringer Ingelheim Investigational Site 133, Heilbronn
  - Boehringer Ingelheim Investigational Site 134, Heilbronn
  - Boehringer Ingelheim Investigational Site 136, Heilbronn
  - Boehringer Ingelheim Investigational Site 139, Heilbronn
  - Boehringer Ingelheim Investigational Site 1216, Heiligenstadt
  - Boehringer Ingelheim Investigational Site 1365, Heilstedt
  - Boehringer Ingelheim Investigational Site 313, Heimstetten
  - Boehringer Ingelheim Investigational Site 636, Heinsberg
  - Boehringer Ingelheim Investigational Site 1142, Heist
  - Boehringer Ingelheim Investigational Site 678, Hellenthal
  - Boehringer Ingelheim Investigational Site 944, Helmstedt
  - Boehringer Ingelheim Investigational Site 946, Helmstedt
  - Boehringer Ingelheim Investigational Site 1071, Hemmoor
  - Boehringer Ingelheim Investigational Site 1072, Hemmoor
  - Boehringer Ingelheim Investigational Site 1076, Hemmoor
  - Boehringer Ingelheim Investigational Site 1078, Hemmoor
  - Boehringer Ingelheim Investigational Site 1498, Hemsbach
  - Boehringer Ingelheim Investigational Site 1499, Hemsbach
  - Boehringer Ingelheim Investigational Site 665, Hennef (Sieg)
  - Boehringer Ingelheim Investigational Site 669, Hennef (Sieg)
  - Boehringer Ingelheim Investigational Site 1334, Hennickendorf
  - Boehringer Ingelheim Investigational Site 1117, Hensted-Ulzburg
  - Boehringer Ingelheim Investigational Site 387, Henstedt-Ulzburg
  - Boehringer Ingelheim Investigational Site 412, Henstedt-Ulzburg
  - Boehringer Ingelheim Investigational Site 1209, Herbsleben
  - Boehringer Ingelheim Investigational Site 873, Herford
  - Boehringer Ingelheim Investigational Site 877, Herford
  - Boehringer Ingelheim Investigational Site 1521, Herne
  - Boehringer Ingelheim Investigational Site 860, Herne
  - Boehringer Ingelheim Investigational Site 861, Herne
  - Boehringer Ingelheim Investigational Site 37, Herrenberg
  - Boehringer Ingelheim Investigational Site 60, Herrenberg-Affstaett
  - Boehringer Ingelheim Investigational Site 1436, Herrnhut
  - Boehringer Ingelheim Investigational Site 162, Heubach
  - Boehringer Ingelheim Investigational Site 617, Heusweiler
  - Boehringer Ingelheim Investigational Site 620, Heusweiler
  - Boehringer Ingelheim Investigational Site 902, Hilden
  - Boehringer Ingelheim Investigational Site 960, Hildesheim
  - Boehringer Ingelheim Investigational Site 217, Hilpoltstein
  - Boehringer Ingelheim Investigational Site 1491, Hirschaid
  - Boehringer Ingelheim Investigational Site 284, Hirschaid
  - Boehringer Ingelheim Investigational Site 364, Hirschau
  - Boehringer Ingelheim Investigational Site 483, Hochheim am Main
  - Boehringer Ingelheim Investigational Site 1313, Hohen Neuendorf/OT Bergfelde
  - Boehringer Ingelheim Investigational Site 372, Hohenau
  - Boehringer Ingelheim Investigational Site 955, Hohenhameln
  - Boehringer Ingelheim Investigational Site 1298, Hohenleipisch
  - Boehringer Ingelheim Investigational Site 1151, Hoisdorf
  - Boehringer Ingelheim Investigational Site 1114, Holm
  - Boehringer Ingelheim Investigational Site 47, Horb
  - Boehringer Ingelheim Investigational Site 1435, Hoyerswerda
  - Boehringer Ingelheim Investigational Site 186, Höchberg
  - Boehringer Ingelheim Investigational Site 187, Höchberg
  - Boehringer Ingelheim Investigational Site 1369, Hötensleben
  - Boehringer Ingelheim Investigational Site 1027, Hude/Wuesting
  - Boehringer Ingelheim Investigational Site 404, Hummeltal
  - Boehringer Ingelheim Investigational Site 657, Hückelhoven
  - Boehringer Ingelheim Investigational Site 667, Hürth
  - Boehringer Ingelheim Investigational Site 851, Ibbenbueren-Dickenberg
  - Boehringer Ingelheim Investigational Site 335, Ichenhausen
  - Boehringer Ingelheim Investigational Site 451, Idar-Oberstein
  - Boehringer Ingelheim Investigational Site 1574, Ifta
  - Boehringer Ingelheim Investigational Site 496, Ingelheim
  - Boehringer Ingelheim Investigational Site 138, Ingersheim
  - Boehringer Ingelheim Investigational Site 196, Ingolstadt
  - Boehringer Ingelheim Investigational Site 214, Ingolstadt
  - Boehringer Ingelheim Investigational Site 215, Ingolstadt
  - Boehringer Ingelheim Investigational Site 285, Ingolstadt
  - Boehringer Ingelheim Investigational Site 621, Irsch/Saar
  - Boehringer Ingelheim Investigational Site 787, Iserlohn
  - Boehringer Ingelheim Investigational Site 331, Ismaning
  - Boehringer Ingelheim Investigational Site 711, Issum
  - Boehringer Ingelheim Investigational Site 1255, Jahnsdorf/Erzgeb.
  - Boehringer Ingelheim Investigational Site 1234, Jena
  - Boehringer Ingelheim Investigational Site 1248, Jena
  - Boehringer Ingelheim Investigational Site 1249, Jena-Lobeda
  - Boehringer Ingelheim Investigational Site 63, Jettingen-Unterjettingen
  - Boehringer Ingelheim Investigational Site 206, Johannesberg
  - Boehringer Ingelheim Investigational Site 1132, Jübek
  - Boehringer Ingelheim Investigational Site 712, Jüchen
  - Boehringer Ingelheim Investigational Site 1609, Jülich
  - Boehringer Ingelheim Investigational Site 623, Jülich
  - Boehringer Ingelheim Investigational Site 607, Jünkerath
  - Boehringer Ingelheim Investigational Site 1424, Kaebschuetztal/OT Kroegis
  - Boehringer Ingelheim Investigational Site 204, Kahl am Main
  - Boehringer Ingelheim Investigational Site 1610, Kaiserslautern
  - Boehringer Ingelheim Investigational Site 422, Kaiserslautern
  - Boehringer Ingelheim Investigational Site 423, Kaiserslautern
  - Boehringer Ingelheim Investigational Site 424, Kaiserslautern
  - Boehringer Ingelheim Investigational Site 430, Kaiserslautern
  - Boehringer Ingelheim Investigational Site 433, Kaiserslautern
  - Boehringer Ingelheim Investigational Site 710, Kalkar
  - Boehringer Ingelheim Investigational Site 811, Kamen
  - Boehringer Ingelheim Investigational Site 815, Kamen
  - Boehringer Ingelheim Investigational Site 758, Kamp-Lintfort
  - Boehringer Ingelheim Investigational Site 1131, Kappeln
  - Boehringer Ingelheim Investigational Site 1593, Karlsruhe
  - Boehringer Ingelheim Investigational Site 1594, Karlsruhe
  - Boehringer Ingelheim Investigational Site 1595, Karlsruhe
  - Boehringer Ingelheim Investigational Site 15, Karlsruhe
  - Boehringer Ingelheim Investigational Site 16, Karlsruhe
  - Boehringer Ingelheim Investigational Site 17, Karlsruhe
  - Boehringer Ingelheim Investigational Site 2, Karlsruhe
  - Boehringer Ingelheim Investigational Site 14, Karlsruhe (Durlach)
  - Boehringer Ingelheim Investigational Site 1551, Kassel
  - Boehringer Ingelheim Investigational Site 1552, Kassel
  - Boehringer Ingelheim Investigational Site 1553, Kassel
  - Boehringer Ingelheim Investigational Site 1554, Kassel
  - Boehringer Ingelheim Investigational Site 1555, Kassel
  - Boehringer Ingelheim Investigational Site 565, Kassel
  - Boehringer Ingelheim Investigational Site 566, Kassel
  - Boehringer Ingelheim Investigational Site 568, Kassel
  - Boehringer Ingelheim Investigational Site 705, Kempen
  - Boehringer Ingelheim Investigational Site 229, Kempten
  - Boehringer Ingelheim Investigational Site 230, Kempten
  - Boehringer Ingelheim Investigational Site 231, Kempten
  - Boehringer Ingelheim Investigational Site 31, Kenzingen
  - Boehringer Ingelheim Investigational Site 501, Kiedrich
  - Boehringer Ingelheim Investigational Site 1101, Kiel
  - Boehringer Ingelheim Investigational Site 1102, Kiel
  - Boehringer Ingelheim Investigational Site 1129, Kiel
  - Boehringer Ingelheim Investigational Site 791, Kierspe
  - Boehringer Ingelheim Investigational Site 30, Kippenheim
  - Boehringer Ingelheim Investigational Site 144, Kirchardt
  - Boehringer Ingelheim Investigational Site 145, Kirchardt
  - Boehringer Ingelheim Investigational Site 365, Kirchenlamitz
  - Boehringer Ingelheim Investigational Site 1208, Kirchheilingen
  - Boehringer Ingelheim Investigational Site 435, Kirchheimbolanden
  - Boehringer Ingelheim Investigational Site 437, Kirchheimbolanden
  - Boehringer Ingelheim Investigational Site 5, Kirchzarten
  - Boehringer Ingelheim Investigational Site 1378, Kleinmachnow
  - Boehringer Ingelheim Investigational Site 1608, Kleinostheim
  - Boehringer Ingelheim Investigational Site 56, Klettgau-Griessen
  - Boehringer Ingelheim Investigational Site 704, Kleve
  - Boehringer Ingelheim Investigational Site 203, Klingenberg
  - Boehringer Ingelheim Investigational Site 1264, Klingenthal
  - Boehringer Ingelheim Investigational Site 648, Koeln (Bilderstoeckchen)
  - Boehringer Ingelheim Investigational Site 676, Koeln-Hoehenberg
  - Boehringer Ingelheim Investigational Site 632, Koeln-Junkersdorf
  - Boehringer Ingelheim Investigational Site 650, Koeln-Lindenthal
  - Boehringer Ingelheim Investigational Site 714, Korschenbroich
  - Boehringer Ingelheim Investigational Site 334, Königsbrunn
  - Boehringer Ingelheim Investigational Site 1412, Königsbrück
  - Boehringer Ingelheim Investigational Site 1342, Köthen
  - Boehringer Ingelheim Investigational Site 1372, Köthen
  - Boehringer Ingelheim Investigational Site 691, Krefeld
  - Boehringer Ingelheim Investigational Site 696, Krefeld
  - Boehringer Ingelheim Investigational Site 706, Krefeld
  - Boehringer Ingelheim Investigational Site 709, Krefeld
  - Boehringer Ingelheim Investigational Site 767, Kreuztal
  - Boehringer Ingelheim Investigational Site 401, Kronach
  - Boehringer Ingelheim Investigational Site 539, Kronberg/Ts.
  - Boehringer Ingelheim Investigational Site 538, Kronberg/Ts
  - Boehringer Ingelheim Investigational Site 1159, Kronshagen
  - Boehringer Ingelheim Investigational Site 1160, Kronshagen
  - Boehringer Ingelheim Investigational Site 325, Krumbach
  - Boehringer Ingelheim Investigational Site 353, Künzing
  - Boehringer Ingelheim Investigational Site 38, L.-Echterdingen
  - Boehringer Ingelheim Investigational Site 367, Laaber
  - Boehringer Ingelheim Investigational Site 1176, Laage
  - Boehringer Ingelheim Investigational Site 1004, Laatzen
  - Boehringer Ingelheim Investigational Site 1124, Laboe
  - Boehringer Ingelheim Investigational Site 541, Lahnau
  - Boehringer Ingelheim Investigational Site 89, Laichingen
  - Boehringer Ingelheim Investigational Site 1191, Lalendorf
  - Boehringer Ingelheim Investigational Site 388, Lampertheim
  - Boehringer Ingelheim Investigational Site 492, Lampertheim
  - Boehringer Ingelheim Investigational Site 510, Lampertheim
  - Boehringer Ingelheim Investigational Site 514, Lampertheim
  - Boehringer Ingelheim Investigational Site 419, Landau
  - Boehringer Ingelheim Investigational Site 1588, Landesbergen
  - Boehringer Ingelheim Investigational Site 322, Landshut
  - Boehringer Ingelheim Investigational Site 90, Langenau
  - Boehringer Ingelheim Investigational Site 915, Langenfeld
  - Boehringer Ingelheim Investigational Site 1001, Langenhagen
  - Boehringer Ingelheim Investigational Site 470, Langenlonsheim
  - Boehringer Ingelheim Investigational Site 1276, Lankwitz
  - Boehringer Ingelheim Investigational Site 1165, Lauenburg
  - Boehringer Ingelheim Investigational Site 384, Lauf
  - Boehringer Ingelheim Investigational Site 1221, Lauscha
  - Boehringer Ingelheim Investigational Site 583, Lauterbach
  - Boehringer Ingelheim Investigational Site 1513, Lähden
  - Boehringer Ingelheim Investigational Site 1332, Lebus
  - Boehringer Ingelheim Investigational Site 1128, Leck
  - Boehringer Ingelheim Investigational Site 1015, Leer
  - Boehringer Ingelheim Investigational Site 1562, Leer
  - Boehringer Ingelheim Investigational Site 982, Lehrte
  - Boehringer Ingelheim Investigational Site 254, Leiblfing
  - Boehringer Ingelheim Investigational Site 44, Leinfelden-Echterdingen
  - Boehringer Ingelheim Investigational Site 329, Leipheim
  - Boehringer Ingelheim Investigational Site 1455, Leipzig
  - Boehringer Ingelheim Investigational Site 1458, Leipzig
  - Boehringer Ingelheim Investigational Site 1462, Leipzig
  - Boehringer Ingelheim Investigational Site 1463, Leipzig
  - Boehringer Ingelheim Investigational Site 1464, Leipzig
  - Boehringer Ingelheim Investigational Site 1465, Leipzig
  - Boehringer Ingelheim Investigational Site 1467, Leipzig
  - Boehringer Ingelheim Investigational Site 1470, Leipzig
  - Boehringer Ingelheim Investigational Site 1471, Leipzig
  - Boehringer Ingelheim Investigational Site 1472, Leipzig
  - Boehringer Ingelheim Investigational Site 1479, Leipzig
  - Boehringer Ingelheim Investigational Site 1516, Leipzig
  - Boehringer Ingelheim Investigational Site 1600, Leipzig
  - Boehringer Ingelheim Investigational Site 1022, Lemwerder
  - Boehringer Ingelheim Investigational Site 1616, Lengede-Woltwiesche
  - Boehringer Ingelheim Investigational Site 956, Lengede-Woltwiesche
  - Boehringer Ingelheim Investigational Site 831, Lengerich
  - Boehringer Ingelheim Investigational Site 835, Lengerich
  - Boehringer Ingelheim Investigational Site 911, Leverkusen
  - Boehringer Ingelheim Investigational Site 920, Leverkusen
  - Boehringer Ingelheim Investigational Site 921, Leverkusen
  - Boehringer Ingelheim Investigational Site 406, Lichtenfels
  - Boehringer Ingelheim Investigational Site 1251, Lichtentanne
  - Boehringer Ingelheim Investigational Site 577, Liebenau
  - Boehringer Ingelheim Investigational Site 833, Lienen-Kattenvenne
  - Boehringer Ingelheim Investigational Site 848, Lienen-Kattenvenne
  - Boehringer Ingelheim Investigational Site 1047, Lilienthal
  - Boehringer Ingelheim Investigational Site 425, Limburgerhof
  - Boehringer Ingelheim Investigational Site 429, Limburgerhof
  - Boehringer Ingelheim Investigational Site 976, Lindhorst
  - Boehringer Ingelheim Investigational Site 983, Lindhorst
  - Boehringer Ingelheim Investigational Site 663, Lindlar
  - Boehringer Ingelheim Investigational Site 664, Lindlar
  - Boehringer Ingelheim Investigational Site 652, Linnich
  - Boehringer Ingelheim Investigational Site 9, Loerrach
  - Boehringer Ingelheim Investigational Site 574, Lohfelden
  - Boehringer Ingelheim Investigational Site 589, Lollar
  - Boehringer Ingelheim Investigational Site 590, Londorf
  - Boehringer Ingelheim Investigational Site 1029, Löhne
  - Boehringer Ingelheim Investigational Site 440, Lu.-Ruchheim
  - Boehringer Ingelheim Investigational Site 1291, Lubin
  - Boehringer Ingelheim Investigational Site 1297, Lubnjow
  - Boehringer Ingelheim Investigational Site 1269, Lucka
  - Boehringer Ingelheim Investigational Site 1290, Luckau
  - Boehringer Ingelheim Investigational Site 1404, Luckenwalde
  - Boehringer Ingelheim Investigational Site 149, Ludwigsburg
  - Boehringer Ingelheim Investigational Site 165, Ludwigsburg
  - Boehringer Ingelheim Investigational Site 173, Ludwigsburg
  - Boehringer Ingelheim Investigational Site 174, Ludwigsburg
  - Boehringer Ingelheim Investigational Site 175, Ludwigsburg
  - Boehringer Ingelheim Investigational Site 181, Ludwigsburg
  - Boehringer Ingelheim Investigational Site 417, Ludwigshafen
  - Boehringer Ingelheim Investigational Site 426, Ludwigshafen
  - Boehringer Ingelheim Investigational Site 1175, Ludwigslust
  - Boehringer Ingelheim Investigational Site 449, Lutzerath
  - Boehringer Ingelheim Investigational Site 1100, Lübeck
  - Boehringer Ingelheim Investigational Site 1120, Lübeck
  - Boehringer Ingelheim Investigational Site 1158, Lübeck
  - Boehringer Ingelheim Investigational Site 772, Lüdenscheid
  - Boehringer Ingelheim Investigational Site 788, Lüdenscheid
  - Boehringer Ingelheim Investigational Site 792, Lüdenscheid
  - Boehringer Ingelheim Investigational Site 793, Lüdenscheid
  - Boehringer Ingelheim Investigational Site 1080, Lüneburg
  - Boehringer Ingelheim Investigational Site 1082, Lüneburg
  - Boehringer Ingelheim Investigational Site 1084, Lüneburg
  - Boehringer Ingelheim Investigational Site 389, Lünen
  - Boehringer Ingelheim Investigational Site 1480, Lützen
  - Boehringer Ingelheim Investigational Site 1184, Lützow
  - Boehringer Ingelheim Investigational Site 1520, Maerkische Heide/ Gross Leuthen
  - Boehringer Ingelheim Investigational Site 1302, Maerkische Heide/Gross Leuthen
  - Boehringer Ingelheim Investigational Site 1341, Magdeburg
  - Boehringer Ingelheim Investigational Site 1347, Magdeburg
  - Boehringer Ingelheim Investigational Site 1525, Magdeburg
  - Boehringer Ingelheim Investigational Site 207, Mainaschaff
  - Boehringer Ingelheim Investigational Site 333, Mainburg
  - Boehringer Ingelheim Investigational Site 481, Mainz
  - Boehringer Ingelheim Investigational Site 482, Mainz
  - Boehringer Ingelheim Investigational Site 485, Mainz
  - Boehringer Ingelheim Investigational Site 487, Mainz
  - Boehringer Ingelheim Investigational Site 493, Mainz
  - Boehringer Ingelheim Investigational Site 494, Mainz
  - Boehringer Ingelheim Investigational Site 495, Mainz
  - Boehringer Ingelheim Investigational Site 500, Mainz
  - Boehringer Ingelheim Investigational Site 32, Malterdingen
  - Boehringer Ingelheim Investigational Site 112, Mannheim
  - Boehringer Ingelheim Investigational Site 115, Mannheim
  - Boehringer Ingelheim Investigational Site 116, Mannheim
  - Boehringer Ingelheim Investigational Site 121, Mannheim
  - Boehringer Ingelheim Investigational Site 124, Mannheim
  - Boehringer Ingelheim Investigational Site 126, Mannheim
  - Boehringer Ingelheim Investigational Site 1529, Mannheim
  - Boehringer Ingelheim Investigational Site 1532, Mannheim
  - Boehringer Ingelheim Investigational Site 123, Mannheim (Almenhof)
  - Boehringer Ingelheim Investigational Site 131, Mannheim (Kaefertal)
  - Boehringer Ingelheim Investigational Site 130, Mannheim (Neuostheim)
  - Boehringer Ingelheim Investigational Site 125, Mannheim (Waldhof)
  - Boehringer Ingelheim Investigational Site 1528, Mannheim (Waldhof)
  - Boehringer Ingelheim Investigational Site 1527, Mannheim-Lindenhof
  - Boehringer Ingelheim Investigational Site 562, Marburg
  - Boehringer Ingelheim Investigational Site 191, Margetshöchheim
  - Boehringer Ingelheim Investigational Site 1453, Markkleeberg
  - Boehringer Ingelheim Investigational Site 1454, Markkleeberg
  - Boehringer Ingelheim Investigational Site 1478, Markkleeberg
  - Boehringer Ingelheim Investigational Site 1266, Markneukirchen
  - Boehringer Ingelheim Investigational Site 208, Marktheidenfeld
  - Boehringer Ingelheim Investigational Site 402, Marktleugast
  - Boehringer Ingelheim Investigational Site 344, Marktredwitz
  - Boehringer Ingelheim Investigational Site 1509, Marl
  - Boehringer Ingelheim Investigational Site 841, Marl
  - Boehringer Ingelheim Investigational Site 854, Marl
  - Boehringer Ingelheim Investigational Site 439, Meckenheim
  - Boehringer Ingelheim Investigational Site 677, Meckenheim
  - Boehringer Ingelheim Investigational Site 410, Meeder
  - Boehringer Ingelheim Investigational Site 690, Meerbusch
  - Boehringer Ingelheim Investigational Site 713, Meerbusch
  - Boehringer Ingelheim Investigational Site 790, Meinerzhagen
  - Boehringer Ingelheim Investigational Site 1231, Meiningen
  - Boehringer Ingelheim Investigational Site 1421, Meissen
  - Boehringer Ingelheim Investigational Site 1445, Meissen
  - Boehringer Ingelheim Investigational Site 1032, Melle
  - Boehringer Ingelheim Investigational Site 1034, Melle
  - Boehringer Ingelheim Investigational Site 558, Melsungen
  - Boehringer Ingelheim Investigational Site 1487, Memmelsdorf-Drosendorf
  - Boehringer Ingelheim Investigational Site 381, Memmelsdorf-Drosendorf
  - Boehringer Ingelheim Investigational Site 784, Menden
  - Boehringer Ingelheim Investigational Site 465, Mendig
  - Boehringer Ingelheim Investigational Site 1447, Merseburg
  - Boehringer Ingelheim Investigational Site 96, Messkirch
  - Boehringer Ingelheim Investigational Site 850, Mettingen
  - Boehringer Ingelheim Investigational Site 71, Metzingen
  - Boehringer Ingelheim Investigational Site 385, Michelau
  - Boehringer Ingelheim Investigational Site 355, Michelsneukirchen
  - Boehringer Ingelheim Investigational Site 1397, Milower Land
  - Boehringer Ingelheim Investigational Site 1398, Milower Land
  - Boehringer Ingelheim Investigational Site 188, Miltenberg
  - Boehringer Ingelheim Investigational Site 875, Minden
  - Boehringer Ingelheim Investigational Site 879, Minden
  - Boehringer Ingelheim Investigational Site 888, Minden
  - Boehringer Ingelheim Investigational Site 889, Minden
  - Boehringer Ingelheim Investigational Site 892, Minden
  - Boehringer Ingelheim Investigational Site 897, Minden
  - Boehringer Ingelheim Investigational Site 1020, Mittegroßefehn
  - Boehringer Ingelheim Investigational Site 1446, Mittweida
  - Boehringer Ingelheim Investigational Site 732, Moers
  - Boehringer Ingelheim Investigational Site 735, Moers
  - Boehringer Ingelheim Investigational Site 759, Moers
  - Boehringer Ingelheim Investigational Site 1138, Molfsee
  - Boehringer Ingelheim Investigational Site 913, Monheim
  - Boehringer Ingelheim Investigational Site 1017, Moormerland
  - Boehringer Ingelheim Investigational Site 1021, Moormerland
  - Boehringer Ingelheim Investigational Site 110, Mosbach
  - Boehringer Ingelheim Investigational Site 111, Mosbach
  - Boehringer Ingelheim Investigational Site 701, Mönchengladbach
  - Boehringer Ingelheim Investigational Site 702, Mönchengladbach
  - Boehringer Ingelheim Investigational Site 718, Mönchengladbach
  - Boehringer Ingelheim Investigational Site 719, Mönchengladbach
  - Boehringer Ingelheim Investigational Site 720, Mönchengladbach
  - Boehringer Ingelheim Investigational Site 721, Mönchengladbach
  - Boehringer Ingelheim Investigational Site 46, Mössingen
  - Boehringer Ingelheim Investigational Site 1576, Muehlhausen/Thuer.
  - Boehringer Ingelheim Investigational Site 82, Munderkingen
  - Boehringer Ingelheim Investigational Site 180, Murrhardt
  - Boehringer Ingelheim Investigational Site 1534, Mühlacker
  - Boehringer Ingelheim Investigational Site 286, Mühldorf
  - Boehringer Ingelheim Investigational Site 314, Mühldorf
  - Boehringer Ingelheim Investigational Site 1205, Mühlhausen
  - Boehringer Ingelheim Investigational Site 1218, Mühlhausen
  - Boehringer Ingelheim Investigational Site 1577, Mühlhausen
  - Boehringer Ingelheim Investigational Site 1586, Mühlhausen
  - Boehringer Ingelheim Investigational Site 1497, Mülheim
  - Boehringer Ingelheim Investigational Site 753, Mülheim
  - Boehringer Ingelheim Investigational Site 755, Mülheim
  - Boehringer Ingelheim Investigational Site 757, Mülheim
  - Boehringer Ingelheim Investigational Site 407, Münchberg
  - Boehringer Ingelheim Investigational Site 242, München
  - Boehringer Ingelheim Investigational Site 243, München
  - Boehringer Ingelheim Investigational Site 258, München
  - Boehringer Ingelheim Investigational Site 260, München
  - Boehringer Ingelheim Investigational Site 261, München
  - Boehringer Ingelheim Investigational Site 262, München
  - Boehringer Ingelheim Investigational Site 265, München
  - Boehringer Ingelheim Investigational Site 266, München
  - Boehringer Ingelheim Investigational Site 267, München
  - Boehringer Ingelheim Investigational Site 278, München
  - Boehringer Ingelheim Investigational Site 279, München
  - Boehringer Ingelheim Investigational Site 280, München
  - Boehringer Ingelheim Investigational Site 283, München
  - Boehringer Ingelheim Investigational Site 287, München
  - Boehringer Ingelheim Investigational Site 288, München
  - Boehringer Ingelheim Investigational Site 289, München
  - Boehringer Ingelheim Investigational Site 290, München
  - Boehringer Ingelheim Investigational Site 291, München
  - Boehringer Ingelheim Investigational Site 294, München
  - Boehringer Ingelheim Investigational Site 297, München
  - Boehringer Ingelheim Investigational Site 298, München
  - Boehringer Ingelheim Investigational Site 310, München
  - Boehringer Ingelheim Investigational Site 311, München
  - Boehringer Ingelheim Investigational Site 312, München
  - Boehringer Ingelheim Investigational Site 316, München
  - Boehringer Ingelheim Investigational Site 318, München
  - Boehringer Ingelheim Investigational Site 319, München
  - Boehringer Ingelheim Investigational Site 320, München
  - Boehringer Ingelheim Investigational Site 321, München
  - Boehringer Ingelheim Investigational Site 332, München
  - Boehringer Ingelheim Investigational Site 869, Münster
  - Boehringer Ingelheim Investigational Site 872, Münster
  - Boehringer Ingelheim Investigational Site 619, Nalbach
  - Boehringer Ingelheim Investigational Site 475, Nassau
  - Boehringer Ingelheim Investigational Site 1394, Nauen
  - Boehringer Ingelheim Investigational Site 160, Nauenstadt
  - Boehringer Ingelheim Investigational Site 379, Nbg.
  - Boehringer Ingelheim Investigational Site 307, Nersingen
  - Boehringer Ingelheim Investigational Site 309, Nersingen
  - Boehringer Ingelheim Investigational Site 679, Nettersheim
  - Boehringer Ingelheim Investigational Site 687, Nettersheim
  - Boehringer Ingelheim Investigational Site 707, Nettetal
  - Boehringer Ingelheim Investigational Site 308, Neu-Ulm
  - Boehringer Ingelheim Investigational Site 328, Neu-Ulm
  - Boehringer Ingelheim Investigational Site 330, Neu-Ulm
  - Boehringer Ingelheim Investigational Site 234, Neubiberg
  - Boehringer Ingelheim Investigational Site 1179, Neubrandenburg
  - Boehringer Ingelheim Investigational Site 1181, Neubrandenburg
  - Boehringer Ingelheim Investigational Site 195, Neuburg am Inn
  - Boehringer Ingelheim Investigational Site 218, Neuburg am Inn
  - Boehringer Ingelheim Investigational Site 183, Neudenau
  - Boehringer Ingelheim Investigational Site 58, Neuhausen ob Eck
  - Boehringer Ingelheim Investigational Site 1557, Neuhof
  - Boehringer Ingelheim Investigational Site 579, Neuhof
  - Boehringer Ingelheim Investigational Site 358, Neukirchen Hl. Blut
  - Boehringer Ingelheim Investigational Site 1135, Neumünster
  - Boehringer Ingelheim Investigational Site 1139, Neumünster
  - Boehringer Ingelheim Investigational Site 1140, Neumünster
  - Boehringer Ingelheim Investigational Site 594, Neunkirchen
  - Boehringer Ingelheim Investigational Site 245, Neuried
  - Boehringer Ingelheim Investigational Site 1401, Neuruppin
  - Boehringer Ingelheim Investigational Site 699, Neuss
  - Boehringer Ingelheim Investigational Site 722, Neuss
  - Boehringer Ingelheim Investigational Site 723, Neuss
  - Boehringer Ingelheim Investigational Site 724, Neuss-Holzheim
  - Boehringer Ingelheim Investigational Site 1115, Neustadt
  - Boehringer Ingelheim Investigational Site 581, Neustadt
  - Boehringer Ingelheim Investigational Site 582, Neustadt
  - Boehringer Ingelheim Investigational Site 975, Neustadt
  - Boehringer Ingelheim Investigational Site 414, Neustadt/Weinstrasse
  - Boehringer Ingelheim Investigational Site 369, Neutraubling
  - Boehringer Ingelheim Investigational Site 452, Neuwied
  - Boehringer Ingelheim Investigational Site 1503, Niederkassel-Rheidt
  - Boehringer Ingelheim Investigational Site 672, Niederkassel-Rheidt
  - Boehringer Ingelheim Investigational Site 970, Niedernwöhren
  - Boehringer Ingelheim Investigational Site 991, Niedernwöhren
  - Boehringer Ingelheim Investigational Site 468, Niederwoerresbach
  - Boehringer Ingelheim Investigational Site 1566, Nienburg
  - Boehringer Ingelheim Investigational Site 995, Nienburg
  - Boehringer Ingelheim Investigational Site 1167, Norderstedt
  - Boehringer Ingelheim Investigational Site 1169, Norderstedt
  - Boehringer Ingelheim Investigational Site 1584, Nordhausen
  - Boehringer Ingelheim Investigational Site 135, Nordheim
  - Boehringer Ingelheim Investigational Site 845, Nordwalde
  - Boehringer Ingelheim Investigational Site 933, Northeim
  - Boehringer Ingelheim Investigational Site 1409, Nossen
  - Boehringer Ingelheim Investigational Site 1423, Nossen
  - Boehringer Ingelheim Investigational Site 216, Nördlingen
  - Boehringer Ingelheim Investigational Site 1483, Nuremberg
  - Boehringer Ingelheim Investigational Site 1484, Nuremberg
  - Boehringer Ingelheim Investigational Site 1601, Nuremberg
  - Boehringer Ingelheim Investigational Site 374, Nuremberg
  - Boehringer Ingelheim Investigational Site 375, Nuremberg
  - Boehringer Ingelheim Investigational Site 376, Nuremberg
  - Boehringer Ingelheim Investigational Site 382, Nuremberg
  - Boehringer Ingelheim Investigational Site 394, Nuremberg
  - Boehringer Ingelheim Investigational Site 395, Nuremberg
  - Boehringer Ingelheim Investigational Site 396, Nuremberg
  - Boehringer Ingelheim Investigational Site 398, Nuremberg
  - Boehringer Ingelheim Investigational Site 399, Nuremberg
  - Boehringer Ingelheim Investigational Site 400, Nuremberg
  - Boehringer Ingelheim Investigational Site 171, Nürtingen
  - Boehringer Ingelheim Investigational Site 509, Ober-Ramstadt
  - Boehringer Ingelheim Investigational Site 1203, Oberdorla
  - Boehringer Ingelheim Investigational Site 1575, Oberdorla
  - Boehringer Ingelheim Investigational Site 728, Oberhausen
  - Boehringer Ingelheim Investigational Site 733, Oberhausen
  - Boehringer Ingelheim Investigational Site 734, Oberhausen
  - Boehringer Ingelheim Investigational Site 754, Oberhausen
  - Boehringer Ingelheim Investigational Site 756, Oberhausen
  - Boehringer Ingelheim Investigational Site 988, Obernkirchen
  - Boehringer Ingelheim Investigational Site 8, Oberried
  - Boehringer Ingelheim Investigational Site 555, Obertshausen-Hausen
  - Boehringer Ingelheim Investigational Site 885, Oelde
  - Boehringer Ingelheim Investigational Site 813, Oer-Erkenschwich
  - Boehringer Ingelheim Investigational Site 1070, Oerel
  - Boehringer Ingelheim Investigational Site 1073, Oerel
  - Boehringer Ingelheim Investigational Site 336, Oettingen in Bayern
  - Boehringer Ingelheim Investigational Site 520, Offenbach
  - Boehringer Ingelheim Investigational Site 525, Offenbach
  - Boehringer Ingelheim Investigational Site 28, Offenburg
  - Boehringer Ingelheim Investigational Site 317, Olching/Neu-Esting
  - Boehringer Ingelheim Investigational Site 1011, Oldenburg
  - Boehringer Ingelheim Investigational Site 1558, Oldenburg
  - Boehringer Ingelheim Investigational Site 1314, Oranienburg
  - Boehringer Ingelheim Investigational Site 1324, Oranienburg
  - Boehringer Ingelheim Investigational Site 1327, Oranienburg
  - Boehringer Ingelheim Investigational Site 1477, Oschatz
  - Boehringer Ingelheim Investigational Site 1515, Oschatz
  - Boehringer Ingelheim Investigational Site 1343, Oschersleben
  - Boehringer Ingelheim Investigational Site 1362, Oschersleben
  - Boehringer Ingelheim Investigational Site 951, Osloß
  - Boehringer Ingelheim Investigational Site 1005, Ostercappeln
  - Boehringer Ingelheim Investigational Site 1591, Osterode
  - Boehringer Ingelheim Investigational Site 965, Osterode
  - Boehringer Ingelheim Investigational Site 85, Ostrach
  - Boehringer Ingelheim Investigational Site 1200, Ostseebad Prerow
  - Boehringer Ingelheim Investigational Site 1199, Ostseeheilbad Zingst
  - Boehringer Ingelheim Investigational Site 1077, Ottendorf
  - Boehringer Ingelheim Investigational Site 432, Otterbach
  - Boehringer Ingelheim Investigational Site 428, Otterstadt
  - Boehringer Ingelheim Investigational Site 239, Ottobrunn bei München
  - Boehringer Ingelheim Investigational Site 256, Ottobrunn bei München
  - Boehringer Ingelheim Investigational Site 804, Paderborn
  - Boehringer Ingelheim Investigational Site 805, Paderborn
  - Boehringer Ingelheim Investigational Site 826, Paderborn
  - Boehringer Ingelheim Investigational Site 1006, Papenburg
  - Boehringer Ingelheim Investigational Site 1007, Papenburg
  - Boehringer Ingelheim Investigational Site 1008, Papenburg
  - Boehringer Ingelheim Investigational Site 1033, Papenburg
  - Boehringer Ingelheim Investigational Site 1039, Papenburg
  - Boehringer Ingelheim Investigational Site 1040, Papenburg
  - Boehringer Ingelheim Investigational Site 1182, Papenburg
  - Boehringer Ingelheim Investigational Site 1505, Papenburg
  - Boehringer Ingelheim Investigational Site 1606, Papenburg
  - Boehringer Ingelheim Investigational Site 1607, Papenburg
  - Boehringer Ingelheim Investigational Site 1183, Parchim
  - Boehringer Ingelheim Investigational Site 349, Passau
  - Boehringer Ingelheim Investigational Site 373, Passau
  - Boehringer Ingelheim Investigational Site 938, Peine
  - Boehringer Ingelheim Investigational Site 939, Peine
  - Boehringer Ingelheim Investigational Site 950, Peine
  - Boehringer Ingelheim Investigational Site 240, Penzberg
  - Boehringer Ingelheim Investigational Site 247, Penzberg
  - Boehringer Ingelheim Investigational Site 268, Penzberg
  - Boehringer Ingelheim Investigational Site 147, Pforzheim
  - Boehringer Ingelheim Investigational Site 1573, Pforzheim
  - Boehringer Ingelheim Investigational Site 50, Pforzheim
  - Boehringer Ingelheim Investigational Site 52, Pforzheim
  - Boehringer Ingelheim Investigational Site 97, Pfullingen
  - Boehringer Ingelheim Investigational Site 513, Pfungstadt
  - Boehringer Ingelheim Investigational Site 416, Pirmasens
  - Boehringer Ingelheim Investigational Site 1416, Pirna
  - Boehringer Ingelheim Investigational Site 1518, Pirna
  - Boehringer Ingelheim Investigational Site 1563, Pirna
  - Boehringer Ingelheim Investigational Site 467, Plaidt
  - Boehringer Ingelheim Investigational Site 272, Planegg
  - Boehringer Ingelheim Investigational Site 351, Plattling
  - Boehringer Ingelheim Investigational Site 1238, Plauen
  - Boehringer Ingelheim Investigational Site 1254, Plauen
  - Boehringer Ingelheim Investigational Site 1265, Plauen
  - Boehringer Ingelheim Investigational Site 324, Pleiskirchen
  - Boehringer Ingelheim Investigational Site 1113, Plön
  - Boehringer Ingelheim Investigational Site 370, Pocking
  - Boehringer Ingelheim Investigational Site 270, Poecking
  - Boehringer Ingelheim Investigational Site 464, Polch
  - Boehringer Ingelheim Investigational Site 1379, Potsdam
  - Boehringer Ingelheim Investigational Site 1380, Potsdam
  - Boehringer Ingelheim Investigational Site 1381, Potsdam
  - Boehringer Ingelheim Investigational Site 1383, Potsdam
  - Boehringer Ingelheim Investigational Site 1393, Potsdam
  - Boehringer Ingelheim Investigational Site 1450, Potsdam
  - Boehringer Ingelheim Investigational Site 1451, Potsdam
  - Boehringer Ingelheim Investigational Site 1452, Potsdam
  - Boehringer Ingelheim Investigational Site 408, Pottenstein
  - Boehringer Ingelheim Investigational Site 1112, Preetz
  - Boehringer Ingelheim Investigational Site 1122, Preetz
  - Boehringer Ingelheim Investigational Site 1399, Premnitz
  - Boehringer Ingelheim Investigational Site 649, Pulheim-Brauweiler
  - Boehringer Ingelheim Investigational Site 271, Pullach
  - Boehringer Ingelheim Investigational Site 1438, Pulsnitz
  - Boehringer Ingelheim Investigational Site 1180, Putbus/Ruegen
  - Boehringer Ingelheim Investigational Site 595, Püttlingen
  - Boehringer Ingelheim Investigational Site 601, Püttlingen
  - Boehringer Ingelheim Investigational Site 1468, Querfurt
  - Boehringer Ingelheim Investigational Site 1428, Radeberg
  - Boehringer Ingelheim Investigational Site 1413, Radebeul
  - Boehringer Ingelheim Investigational Site 910, Radevormwald
  - Boehringer Ingelheim Investigational Site 49, Radolfzell
  - Boehringer Ingelheim Investigational Site 1440, Ralbitz-Rosenthal
  - Boehringer Ingelheim Investigational Site 12, Rastatt
  - Boehringer Ingelheim Investigational Site 11, Rastatt-Wintersdorf
  - Boehringer Ingelheim Investigational Site 441, Raubach
  - Boehringer Ingelheim Investigational Site 107, Ravensburg
  - Boehringer Ingelheim Investigational Site 832, Recke
  - Boehringer Ingelheim Investigational Site 849, Recke
  - Boehringer Ingelheim Investigational Site 839, Recklinghausen
  - Boehringer Ingelheim Investigational Site 343, Regensburg
  - Boehringer Ingelheim Investigational Site 345, Regensburg
  - Boehringer Ingelheim Investigational Site 368, Regensburg
  - Boehringer Ingelheim Investigational Site 930, Remscheid
  - Boehringer Ingelheim Investigational Site 931, Remscheid
  - Boehringer Ingelheim Investigational Site 168, Remseck-Aldingen
  - Boehringer Ingelheim Investigational Site 166, Remseck
  - Boehringer Ingelheim Investigational Site 458, Rennerod
  - Boehringer Ingelheim Investigational Site 150, Reutlingen
  - Boehringer Ingelheim Investigational Site 151, Reutlingen
  - Boehringer Ingelheim Investigational Site 152, Reutlingen
  - Boehringer Ingelheim Investigational Site 170, Reutlingen
  - Boehringer Ingelheim Investigational Site 172, Reutlingen
  - Boehringer Ingelheim Investigational Site 742, Rheinberg
  - Boehringer Ingelheim Investigational Site 35, Rheinmuenster-Schwarzach
  - Boehringer Ingelheim Investigational Site 10, Rheinstetten
  - Boehringer Ingelheim Investigational Site 479, Rieden
  - Boehringer Ingelheim Investigational Site 438, Rieschweiler
  - Boehringer Ingelheim Investigational Site 894, Rietberg-Neuenkirchen
  - Boehringer Ingelheim Investigational Site 967, Rittmarshausen
  - Boehringer Ingelheim Investigational Site 1263, Rodewisch
  - Boehringer Ingelheim Investigational Site 1299, Roederland-Proesen
  - Boehringer Ingelheim Investigational Site 392, Roederland-Proesen
  - Boehringer Ingelheim Investigational Site 1348, Rohrberg
  - Boehringer Ingelheim Investigational Site 1087, Rosengarten
  - Boehringer Ingelheim Investigational Site 249, Rosenheim
  - Boehringer Ingelheim Investigational Site 251, Rosenheim
  - Boehringer Ingelheim Investigational Site 257, Rosenheim
  - Boehringer Ingelheim Investigational Site 1172, Rostock
  - Boehringer Ingelheim Investigational Site 1189, Rostock
  - Boehringer Ingelheim Investigational Site 1060, Rotenburg (Wümme)
  - Boehringer Ingelheim Investigational Site 578, Rotenburg (Wümme)
  - Boehringer Ingelheim Investigational Site 236, Rottach-Weissach
  - Boehringer Ingelheim Investigational Site 1481, Röcknitz
  - Boehringer Ingelheim Investigational Site 553, Rödermark
  - Boehringer Ingelheim Investigational Site 164, Rudersberg
  - Boehringer Ingelheim Investigational Site 671, Ruppichteroth
  - Boehringer Ingelheim Investigational Site 1337, Rüdersdorf
  - Boehringer Ingelheim Investigational Site 598, Saarbrücken
  - Boehringer Ingelheim Investigational Site 605, Saarbrücken
  - Boehringer Ingelheim Investigational Site 616, Saarbrücken
  - Boehringer Ingelheim Investigational Site 618, Saarbrücken
  - Boehringer Ingelheim Investigational Site 597, Saarlouis
  - Boehringer Ingelheim Investigational Site 33, Saint Blasien
  - Boehringer Ingelheim Investigational Site 255, Salching
  - Boehringer Ingelheim Investigational Site 1353, Salzatal/OT Schiepzig
  - Boehringer Ingelheim Investigational Site 1344, Salzatal
  - Boehringer Ingelheim Investigational Site 1345, Salzatal
  - Boehringer Ingelheim Investigational Site 1036, Salzbergen
  - Boehringer Ingelheim Investigational Site 957, Salzgitter (Lebenstedt)
  - Boehringer Ingelheim Investigational Site 959, Salzgitter (Lebenstedt)
  - Boehringer Ingelheim Investigational Site 1359, Salzmünde
  - Boehringer Ingelheim Investigational Site 1360, Salzmünde
  - Boehringer Ingelheim Investigational Site 348, Salzweg Bei Passau
  - Boehringer Ingelheim Investigational Site 383, Sand
  - Boehringer Ingelheim Investigational Site 1166, Sandesneben
  - Boehringer Ingelheim Investigational Site 688, Sankt Augustin
  - Boehringer Ingelheim Investigational Site 141, Sankt Leon-Rot
  - Boehringer Ingelheim Investigational Site 1504, Sarstedt
  - Boehringer Ingelheim Investigational Site 958, Sarstedt
  - Boehringer Ingelheim Investigational Site 411, Schenefeld
  - Boehringer Ingelheim Investigational Site 1202, Schlagsdorf
  - Boehringer Ingelheim Investigational Site 274, Schleching
  - Boehringer Ingelheim Investigational Site 895, Schloss Holte-Stukenbrock
  - Boehringer Ingelheim Investigational Site 1230, Schlotheim
  - Boehringer Ingelheim Investigational Site 1220, Schmalkalden
  - Boehringer Ingelheim Investigational Site 596, Schmelz
  - Boehringer Ingelheim Investigational Site 1261, Schneeberg
  - Boehringer Ingelheim Investigational Site 1201, Schoenberg/Meckl.
  - Boehringer Ingelheim Investigational Site 1517, Schoensee
  - Boehringer Ingelheim Investigational Site 361, Schoensee
  - Boehringer Ingelheim Investigational Site 948, Schoeppenstadt
  - Boehringer Ingelheim Investigational Site 23, Schopfheim
  - Boehringer Ingelheim Investigational Site 27, Schopfheim
  - Boehringer Ingelheim Investigational Site 163, Schorndorf
  - Boehringer Ingelheim Investigational Site 176, Schorndorf
  - Boehringer Ingelheim Investigational Site 182, Schorndorf
  - Boehringer Ingelheim Investigational Site 1012, Schortens
  - Boehringer Ingelheim Investigational Site 69, Schömberg
  - Boehringer Ingelheim Investigational Site 1126, Schönberg
  - Boehringer Ingelheim Investigational Site 1361, Schönebeck
  - Boehringer Ingelheim Investigational Site 39, Schramberg-Sulgen
  - Boehringer Ingelheim Investigational Site 61, Schramberg-Sulgen
  - Boehringer Ingelheim Investigational Site 1144, Schriesheim
  - Boehringer Ingelheim Investigational Site 1530, Schriesheim
  - Boehringer Ingelheim Investigational Site 1531, Schriesheim
  - Boehringer Ingelheim Investigational Site 1533, Schriesheim
  - Boehringer Ingelheim Investigational Site 29, Schutterwald
  - Boehringer Ingelheim Investigational Site 341, Schwabhausen
  - Boehringer Ingelheim Investigational Site 299, Schwaig B. Nbg.
  - Boehringer Ingelheim Investigational Site 1559, Schwarzenbach A. Wald
  - Boehringer Ingelheim Investigational Site 403, Schwarzenbach A. Wald
  - Boehringer Ingelheim Investigational Site 1524, Schwarzenbek
  - Boehringer Ingelheim Investigational Site 1485, Schwarzenbruck
  - Boehringer Ingelheim Investigational Site 153, Schwäbisch Hall
  - Boehringer Ingelheim Investigational Site 1171, Schwerin
  - Boehringer Ingelheim Investigational Site 1173, Schwerin
  - Boehringer Ingelheim Investigational Site 1174, Schwerin
  - Boehringer Ingelheim Investigational Site 1197, Schwerin
  - Boehringer Ingelheim Investigational Site 1535, Schwetzingen
  - Boehringer Ingelheim Investigational Site 1613, Schwetzingen
  - Boehringer Ingelheim Investigational Site 67, Schwieberdingen
  - Boehringer Ingelheim Investigational Site 232, Seeg
  - Boehringer Ingelheim Investigational Site 1333, Seelow
  - Boehringer Ingelheim Investigational Site 1537, Seelow
  - Boehringer Ingelheim Investigational Site 1548, Seelow
  - Boehringer Ingelheim Investigational Site 1003, Sehnde
  - Boehringer Ingelheim Investigational Site 880, Sendenhorst
  - Boehringer Ingelheim Investigational Site 1602, Siegen
  - Boehringer Ingelheim Investigational Site 1603, Siegen
  - Boehringer Ingelheim Investigational Site 1604, Siegen
  - Boehringer Ingelheim Investigational Site 1605, Siegen
  - Boehringer Ingelheim Investigational Site 763, Siegen
  - Boehringer Ingelheim Investigational Site 764, Siegen
  - Boehringer Ingelheim Investigational Site 765, Siegen
  - Boehringer Ingelheim Investigational Site 766, Siegen
  - Boehringer Ingelheim Investigational Site 624, Simmerath
  - Boehringer Ingelheim Investigational Site 469, Simmertal
  - Boehringer Ingelheim Investigational Site 53, Singen
  - Boehringer Ingelheim Investigational Site 571, Soehrewald
  - Boehringer Ingelheim Investigational Site 819, Soest
  - Boehringer Ingelheim Investigational Site 904, Solingen
  - Boehringer Ingelheim Investigational Site 905, Solingen
  - Boehringer Ingelheim Investigational Site 922, Solingen
  - Boehringer Ingelheim Investigational Site 923, Solingen
  - Boehringer Ingelheim Investigational Site 924, Solingen
  - Boehringer Ingelheim Investigational Site 537, Solms
  - Boehringer Ingelheim Investigational Site 1049, Soltau
  - Boehringer Ingelheim Investigational Site 1088, Soltau
  - Boehringer Ingelheim Investigational Site 1210, Sondershausen
  - Boehringer Ingelheim Investigational Site 1214, Sondershausen
  - Boehringer Ingelheim Investigational Site 1226, Sondershausen
  - Boehringer Ingelheim Investigational Site 1585, Sondershausen
  - Boehringer Ingelheim Investigational Site 1227, Sonnenstein
  - Boehringer Ingelheim Investigational Site 708, Sonsbeck
  - Boehringer Ingelheim Investigational Site 1211, Sömmerda
  - Boehringer Ingelheim Investigational Site 210, Spardorf
  - Boehringer Ingelheim Investigational Site 222, Spardorf
  - Boehringer Ingelheim Investigational Site 609, Speicher
  - Boehringer Ingelheim Investigational Site 612, Spiesen-Elversberg
  - Boehringer Ingelheim Investigational Site 613, Spiesen-Elversberg
  - Boehringer Ingelheim Investigational Site 1300, Spremberg
  - Boehringer Ingelheim Investigational Site 1043, Stade
  - Boehringer Ingelheim Investigational Site 1044, Stade
  - Boehringer Ingelheim Investigational Site 1075, Stade
  - Boehringer Ingelheim Investigational Site 978, Stadthagen
  - Boehringer Ingelheim Investigational Site 990, Stadthagen
  - Boehringer Ingelheim Investigational Site 857, Stadtlohn
  - Boehringer Ingelheim Investigational Site 99, Staig
  - Boehringer Ingelheim Investigational Site 1245, Starkenberg
  - Boehringer Ingelheim Investigational Site 1444, Stauchitz
  - Boehringer Ingelheim Investigational Site 591, Staufenberg
  - Boehringer Ingelheim Investigational Site 1492, Stegaurach
  - Boehringer Ingelheim Investigational Site 281, Stegaurach
  - Boehringer Ingelheim Investigational Site 461, Steimel
  - Boehringer Ingelheim Investigational Site 1037, Steinfeld
  - Boehringer Ingelheim Investigational Site 1185, Sternberg
  - Boehringer Ingelheim Investigational Site 59, Stockach
  - Boehringer Ingelheim Investigational Site 645, Stolberg-Vicht
  - Boehringer Ingelheim Investigational Site 1567, Stolzenau
  - Boehringer Ingelheim Investigational Site 996, Stolzenau
  - Boehringer Ingelheim Investigational Site 1561, Stödtlen
  - Boehringer Ingelheim Investigational Site 157, Stödtlen
  - Boehringer Ingelheim Investigational Site 346, Straubing
  - Boehringer Ingelheim Investigational Site 356, Straubing
  - Boehringer Ingelheim Investigational Site 1317, Strausberg
  - Boehringer Ingelheim Investigational Site 972, Stuhr OT Brinkum
  - Boehringer Ingelheim Investigational Site 973, Stuhr OT Brinkum
  - Boehringer Ingelheim Investigational Site 167, Stuttgart
  - Boehringer Ingelheim Investigational Site 70, Stuttgart
  - Boehringer Ingelheim Investigational Site 177, Stuttgart-Untertuerkheim
  - Boehringer Ingelheim Investigational Site 685, Swisttal-Heimerzheim
  - Boehringer Ingelheim Investigational Site 184, Tauberbischofsheim
  - Boehringer Ingelheim Investigational Site 1391, Teltow
  - Boehringer Ingelheim Investigational Site 1187, Teterow
  - Boehringer Ingelheim Investigational Site 1188, Teterow
  - Boehringer Ingelheim Investigational Site 1448, Teuchern
  - Boehringer Ingelheim Investigational Site 1449, Teuchern
  - Boehringer Ingelheim Investigational Site 366, Tirschenreuth
  - Boehringer Ingelheim Investigational Site 1193, Torgelow
  - Boehringer Ingelheim Investigational Site 1198, Torgelow
  - Boehringer Ingelheim Investigational Site 244, Traunreut
  - Boehringer Ingelheim Investigational Site 250, Traunreut
  - Boehringer Ingelheim Investigational Site 277, Traunreut
  - Boehringer Ingelheim Investigational Site 1403, Trebbin
  - Boehringer Ingelheim Investigational Site 1405, Trebbin
  - Boehringer Ingelheim Investigational Site 447, Treis-Karden
  - Boehringer Ingelheim Investigational Site 199, Treuchtlingen
  - Boehringer Ingelheim Investigational Site 600, Trier
  - Boehringer Ingelheim Investigational Site 622, Trier
  - Boehringer Ingelheim Investigational Site 1177, Tutow
  - Boehringer Ingelheim Investigational Site 45, Tübingen
  - Boehringer Ingelheim Investigational Site 1486, Uchte
  - Boehringer Ingelheim Investigational Site 1568, Uchte
  - Boehringer Ingelheim Investigational Site 1081, Uelzen
  - Boehringer Ingelheim Investigational Site 100, Ulm
  - Boehringer Ingelheim Investigational Site 101, Ulm
  - Boehringer Ingelheim Investigational Site 73, Ulm
  - Boehringer Ingelheim Investigational Site 74, Ulm
  - Boehringer Ingelheim Investigational Site 75, Ulm
  - Boehringer Ingelheim Investigational Site 1560, Unterschneidheim
  - Boehringer Ingelheim Investigational Site 386, Untersiemau
  - Boehringer Ingelheim Investigational Site 614, Urexweiler
  - Boehringer Ingelheim Investigational Site 644, Übach-Palenberg
  - Boehringer Ingelheim Investigational Site 1031, Vechta
  - Boehringer Ingelheim Investigational Site 1035, Vechta-Langfoerden
  - Boehringer Ingelheim Investigational Site 916, Velbert
  - Boehringer Ingelheim Investigational Site 564, Vellmar
  - Boehringer Ingelheim Investigational Site 576, Vellmar
  - Boehringer Ingelheim Investigational Site 992, Verden an der Aller
  - Boehringer Ingelheim Investigational Site 1273, Vetschau
  - Boehringer Ingelheim Investigational Site 1293, Vetschau
  - Boehringer Ingelheim Investigational Site 1295, Vetschau
  - Boehringer Ingelheim Investigational Site 1493, Viereth
  - Boehringer Ingelheim Investigational Site 515, Viernheim
  - Boehringer Ingelheim Investigational Site 604, VK-Fuerstenhausen
  - Boehringer Ingelheim Investigational Site 202, Vohburg an der Donau
  - Boehringer Ingelheim Investigational Site 66, Vöhrenbach
  - Boehringer Ingelheim Investigational Site 606, Völklingen
  - Boehringer Ingelheim Investigational Site 62, VS-Schwenningen
  - Boehringer Ingelheim Investigational Site 64, VS-Villingen
  - Boehringer Ingelheim Investigational Site 65, VS-Villingen
  - Boehringer Ingelheim Investigational Site 155, Waiblingen
  - Boehringer Ingelheim Investigational Site 459, Waldbreitbach
  - Boehringer Ingelheim Investigational Site 572, Waldkappel
  - Boehringer Ingelheim Investigational Site 503, Walluf
  - Boehringer Ingelheim Investigational Site 974, Walsrode
  - Boehringer Ingelheim Investigational Site 1019, Wangerland
  - Boehringer Ingelheim Investigational Site 829, Warburg
  - Boehringer Ingelheim Investigational Site 1009, Wardenburg
  - Boehringer Ingelheim Investigational Site 1508, Wardenburg
  - Boehringer Ingelheim Investigational Site 390, Wardenburg
  - Boehringer Ingelheim Investigational Site 870, Warendorf
  - Boehringer Ingelheim Investigational Site 808, Warstein
  - Boehringer Ingelheim Investigational Site 827, Warstein
  - Boehringer Ingelheim Investigational Site 105, Warthausen
  - Boehringer Ingelheim Investigational Site 628, Wassenberg
  - Boehringer Ingelheim Investigational Site 640, Wassenberg
  - Boehringer Ingelheim Investigational Site 545, Wächtersbach
  - Boehringer Ingelheim Investigational Site 103, Wäschenbeuren
  - Boehringer Ingelheim Investigational Site 1141, Wedel
  - Boehringer Ingelheim Investigational Site 658, Wegberg
  - Boehringer Ingelheim Investigational Site 653, Wegberg-Beeck
  - Boehringer Ingelheim Investigational Site 462, Weibern
  - Boehringer Ingelheim Investigational Site 22, Weil am Rhein
  - Boehringer Ingelheim Investigational Site 1206, Weinbergen OT Bollstedt
  - Boehringer Ingelheim Investigational Site 1578, Weinbergen OT Bollstedt
  - Boehringer Ingelheim Investigational Site 114, Weinheim
  - Boehringer Ingelheim Investigational Site 119, Weinheim
  - Boehringer Ingelheim Investigational Site 179, Weissach I. T.
  - Boehringer Ingelheim Investigational Site 1228, Weissensee
  - Boehringer Ingelheim Investigational Site 463, Weißenthurm
  - Boehringer Ingelheim Investigational Site 909, Wermelskirchen
  - Boehringer Ingelheim Investigational Site 1473, Wermsdorf
  - Boehringer Ingelheim Investigational Site 1474, Wermsdorf
  - Boehringer Ingelheim Investigational Site 1475, Wermsdorf
  - Boehringer Ingelheim Investigational Site 391, Wermsdorf
  - Boehringer Ingelheim Investigational Site 1363, Wernigerode
  - Boehringer Ingelheim Investigational Site 1364, Wernigerode
  - Boehringer Ingelheim Investigational Site 1367, Wernigerode
  - Boehringer Ingelheim Investigational Site 161, Wertheim am Main
  - Boehringer Ingelheim Investigational Site 855, Wesel
  - Boehringer Ingelheim Investigational Site 856, Wesel
  - Boehringer Ingelheim Investigational Site 681, Wesseling
  - Boehringer Ingelheim Investigational Site 846, Westerkappeln
  - Boehringer Ingelheim Investigational Site 587, Wetter
  - Boehringer Ingelheim Investigational Site 1512, Wetzlar
  - Boehringer Ingelheim Investigational Site 455, Wetzlar
  - Boehringer Ingelheim Investigational Site 519, Wetzlar
  - Boehringer Ingelheim Investigational Site 523, Wetzlar
  - Boehringer Ingelheim Investigational Site 536, Wetzlar
  - Boehringer Ingelheim Investigational Site 540, Wetzlar-Dutenhofen
  - Boehringer Ingelheim Investigational Site 1178, Weyhe
  - Boehringer Ingelheim Investigational Site 1569, Weyhe
  - Boehringer Ingelheim Investigational Site 969, Weyhe
  - Boehringer Ingelheim Investigational Site 993, Weyhe
  - Boehringer Ingelheim Investigational Site 994, Weyhe
  - Boehringer Ingelheim Investigational Site 997, Weyhe
  - Boehringer Ingelheim Investigational Site 998, Weyhe OT Leeste
  - Boehringer Ingelheim Investigational Site 1570, Weyhe OT Mitte
  - Boehringer Ingelheim Investigational Site 817, Wickede/Ruhr
  - Boehringer Ingelheim Investigational Site 480, Wiesbaden
  - Boehringer Ingelheim Investigational Site 484, Wiesbaden
  - Boehringer Ingelheim Investigational Site 486, Wiesbaden
  - Boehringer Ingelheim Investigational Site 491, Wiesbaden
  - Boehringer Ingelheim Investigational Site 502, Wiesbaden
  - Boehringer Ingelheim Investigational Site 505, Wiesbaden
  - Boehringer Ingelheim Investigational Site 506, Wiesbaden
  - Boehringer Ingelheim Investigational Site 507, Wiesbaden
  - Boehringer Ingelheim Investigational Site 508, Wiesbaden
  - Boehringer Ingelheim Investigational Site 109, Wiesloch
  - Boehringer Ingelheim Investigational Site 1536, Wiesloch
  - Boehringer Ingelheim Investigational Site 1000, Wietzen
  - Boehringer Ingelheim Investigational Site 1016, Wilhelmshaven
  - Boehringer Ingelheim Investigational Site 1041, Wilhelmshaven
  - Boehringer Ingelheim Investigational Site 1042, Wilhelmshaven
  - Boehringer Ingelheim Investigational Site 1013, Wilhelmshaven-Voslapp
  - Boehringer Ingelheim Investigational Site 703, Willich
  - Boehringer Ingelheim Investigational Site 359, Windischeschenbach
  - Boehringer Ingelheim Investigational Site 360, Windischeschenbach
  - Boehringer Ingelheim Investigational Site 1086, Winsen
  - Boehringer Ingelheim Investigational Site 984, Winsen
  - Boehringer Ingelheim Investigational Site 928, Wipperfürth
  - Boehringer Ingelheim Investigational Site 929, Wipperfürth
  - Boehringer Ingelheim Investigational Site 770, Witten
  - Boehringer Ingelheim Investigational Site 774, Witten
  - Boehringer Ingelheim Investigational Site 776, Witten
  - Boehringer Ingelheim Investigational Site 1459, Wittenberg
  - Boehringer Ingelheim Investigational Site 1469, Wittenberg
  - Boehringer Ingelheim Investigational Site 1402, Wittenberge
  - Boehringer Ingelheim Investigational Site 602, Wittlich
  - Boehringer Ingelheim Investigational Site 608, Wittlich
  - Boehringer Ingelheim Investigational Site 610, Wittlich
  - Boehringer Ingelheim Investigational Site 1018, Wittmund
  - Boehringer Ingelheim Investigational Site 1400, Wittstock
  - Boehringer Ingelheim Investigational Site 575, Witzenhausen
  - Boehringer Ingelheim Investigational Site 1571, Wolfenbüttel
  - Boehringer Ingelheim Investigational Site 945, Wolfenbüttel
  - Boehringer Ingelheim Investigational Site 953, Wolfenbüttel
  - Boehringer Ingelheim Investigational Site 263, Wolfratshausen
  - Boehringer Ingelheim Investigational Site 947, Wolfsburg
  - Boehringer Ingelheim Investigational Site 952, Wolfsburg-Reislingen
  - Boehringer Ingelheim Investigational Site 197, Wolnzach
  - Boehringer Ingelheim Investigational Site 497, Wöllstein
  - Boehringer Ingelheim Investigational Site 498, Wöllstein
  - Boehringer Ingelheim Investigational Site 1565, Wunstorf
  - Boehringer Ingelheim Investigational Site 907, Wuppertal
  - Boehringer Ingelheim Investigational Site 912, Wuppertal
  - Boehringer Ingelheim Investigational Site 925, Wuppertal
  - Boehringer Ingelheim Investigational Site 926, Wuppertal
  - Boehringer Ingelheim Investigational Site 927, Wuppertal
  - Boehringer Ingelheim Investigational Site 639, Würselen
  - Boehringer Ingelheim Investigational Site 1286, Zeesen
  - Boehringer Ingelheim Investigational Site 301, Zeil
  - Boehringer Ingelheim Investigational Site 1223, Zella-Mehlis
  - Boehringer Ingelheim Investigational Site 352, Zenting
  - Boehringer Ingelheim Investigational Site 1395, Zernitz-Lohm
  - Boehringer Ingelheim Investigational Site 1287, Zeuthen
  - Boehringer Ingelheim Investigational Site 43, Zimmern
  - Boehringer Ingelheim Investigational Site 357, Zinzenzell
  - Boehringer Ingelheim Investigational Site 397, Zirndorf
  - Boehringer Ingelheim Investigational Site 1419, Zittau
  - Boehringer Ingelheim Investigational Site 1579, Zittau
  - Boehringer Ingelheim Investigational Site 282, Zorneding
  - Boehringer Ingelheim Investigational Site 305, Zusmarshausen
  - Boehringer Ingelheim Investigational Site 421, Zweibrücken
  - Boehringer Ingelheim Investigational Site 1243, Zwickau
  - Boehringer Ingelheim Investigational Site 1244, Zwickau
  - Boehringer Ingelheim Investigational Site 1252, Zwickau

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Reasons for exclusion from analysis: 25 patients were documented as having severe renal impairment (RI), 1643 patients were acc. to documentation either not renally impaired or degree of RI was unknown or missing. Acc. to documentation 120 patients had valvular atrial fibrillation (AF), in 922 patients the origin of AF was unknown or missing.
Pre-assignment Details: 4340 patients were enrolled in the study, 2220 patients had no documented mild or moderate renal impairment or no documented non valvular atrial fibrillation. Therefore, 2120 patients remained for analysis.
Groups:
- All Patients: All patients with documented mild or moderate renal impairment and non valvular atrial fibrillation (Per Protocol Set, PPS).
Period: Overall Study
Arm/Group | All Patients
Started | 2120
Completed | 2120
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All patients with documented mild or moderate renal impairment and non valvular atrial fibrillation (PPS).
Groups:
- All Patients: All patients with documented mild or moderate renal impairment and non valvular atrial fibrillation (PPS).
Arm/Group | All Patients
Number analyzed (Participants) | 2120
Age, Continuous [Mean (Standard Deviation); unit: years] — For 5 patients the documentation of date of birth is missing, so age could be calculated for N=2115 patients.
  years | 75.2 (8.8)
Gender [Number; unit: participants] — For 4 patients the documentation of gender is missing.
  participants
    Female | 1015
    Male | 1101

OUTCOME MEASURES:

1. Primary Outcome: Creatinine Clearance (Recalculated Using Entries of Age, Gender, Body Weight and Serum Creatinine Made by the Physician)
Description: The creatinine clearance was recalculated with the Cockcroft-Gault formula using age, gender, body weight, and serum creatinine.
Time Frame: One single observation time point: at the time of prescription before the first intake of dabigatran etexilate
Population: All patients with documented mild or moderate renal impairment and non-valvular atrial fibrillation (PPS) having evaluable data for age, gender, body weight, and serum creatinine. In 145 patients age, gender, serum creatinine or weight was missing so that Creatinine Clearance according to the Cockcroft Gault formula could not be recalculated.
Measure: Median (Inter-Quartile Range); unit: ml/min
Arm/Group | All Patients
Number analyzed (Participants) | 1975
ml/min | 55.2 [43.6 to 68.3]

ADVERSE EVENTS:
Time Frame: One single observation time point: at the time of prescription before the first intake of dabigatran etexilate
Description: Patients were documented at the time of the first prescription of dabigatran etexilate within the study period and before the first intake of Pradaxa®.
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
This non-interventional studies is conducted according to §67, section 6 German Medicines Act. The term 'principal investigator' is not applicable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes